CLINICAL TRIAL: NCT02831673
Title: A Phase III, Randomised, Double Blind, Multicentre, Parallel Group, Non Inferiority Study Evaluating the Efficacy, Safety, and Tolerability of Dolutegravir Plus Lamivudine Compared to Dolutegravir Plus Tenofovir/Emtricitabine in Human Immunodeficiency Virus 1 Infected Treatment naïve Adults
Brief Title: An Efficacy, Safety, and Tolerability Study Comparing Dolutegravir Plus Lamivudine With Dolutegravir Plus Tenofovir/Emtricitabine in Treatment naïve HIV Infected Subjects (Gemini 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: PPD Development, LP (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204861; 2015-004418-95 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-13 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-07

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: safety; treatment naïve; HIV 1; dolutegravir plus lamivudine; non inferiority; tolerability; dolutegravir plus tenofovir/emtricitabine; efficacy
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir; Lamivudine; Tenofovir; Emtricitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DTG + 3TC (50 mg+300 mg) (Experimental): Eligible participants will receive one 50 mg tablet of DTG plus one overencapsulated 300 mg 3TC tablet orally once daily upto 96 weeks; thereafter will receive DTG plus 3TC tablet upto Week 148 and will continue to receive this schedule until (i) DTG and 3TC are both locally approved for use as part of a dual regimen, and the single entities of DTG and 3TC are available to patients (e.g. through public health services), or (ii) the DTG/3TC FDC tablet, if required by local regulations, is available, , or (iii) the participant no longer derives clinical benefit, or (iv) the participant meets a protocol defined reason for discontinuation, or (v) development of the DTG plus 3TC dual regimen is terminated.
  Interventions: Drug: Dolutegravir (DTG); Drug: Lamivudine (3TC)
- DTG + TDF/FTC FDC (50 mg+300/200 mg) (Active Comparator): Eligible participants will receive one 50 mg tablet of DTG plus one overencapsulated TDF/ FTC FDC (300/200 mg) tablet orally once daily upto 96 weeks; thereafter will receive DTG plus TDF/FTC FDC tablets upto Week 148 (open-label randomised phase).
  Interventions: Drug: Dolutegravir (DTG); Drug: Tenofovir disoproxil fumarate/Emtricitabine (TDF/FTC FDC)

INTERVENTIONS:
Drug: Dolutegravir (DTG) — DTG is available as 50 mg white, round, biconvex, film coated tablet debossed on one side with 'SV 572' and on the other side with '50'. The tablets are packaged into high density polyethylene (HDPE) bottles with induction seals and child resistant closures. Each 45 ml bottle contains 30 tablets and a desiccant. DTG 50 mg tablet will be orally administered once daily with or without food upto 148 weeks.
Drug: Lamivudine (3TC) — Lamivudine is available as swedish orange, 'AA' sized elongated double blind HPMC capsules containing 300 mg lamivudine to visually match overencapsulated TDF/FTC FDC tablet. The capsules are packaged into HDPE bottles with induction seals and child resistant closures. Each 150 mL bottle contains 30 capsules and a desiccant. Overencapsulated 3TC 300 mg tablet will be orally administered once daily with or without food upto 96 weeks. From Week 96 to Week 148, lamivudine will be dispensed as 300 mg white, diamond shaped, scored, film coated tablets debossed with 'GX CJ7' on both sides, packed in over labelled HDPE bottles with child-resistant closures each containing 30 tablets.
  Arms: DTG + 3TC (50 mg+300 mg)
Drug: Tenofovir disoproxil fumarate/Emtricitabine (TDF/FTC FDC) — Tenofovir disoproxil fumarate and Emtricitabine are available as swedish orange, 'AA' sized elongated double blind HPMC capsules containing 300 mg TDF and 200 mg FTC to visually match overencapsulated 3TC tablet. The capsules are packaged into HDPE bottles with induction seals and child resistant closures. Each 150 mL bottle contains 30 capsules and a desiccant. Overencapsulated tenofovir disoproxil fumarate/emtricitabine tablet will be orally administered once daily with or without food upto 96 weeks. From Week 96 to Week 148, tenofovir disoproxil fumarate/emtricitabine will be dispensed as 300/200 mg white, blue, capsule shaped, film coated tablets debossed with 'GILEAD' on one side and '701' on another side, packed in overlabelled HDPE bottles with polypropylene childresistant closures each containing 30 tablets and a desiccant.
  Arms: DTG + TDF/FTC FDC (50 mg+300/200 mg)

SUMMARY:
This study will compare safety, efficacy, and tolerability of a two drug regimen of dolutegravir (DTG) plus (+) lamivudine (3TC) administered once daily with DTG plus two nucleoside reverse transcriptase inhibitors (Tenofovir [TDF]/Emtricitabine [FTC] fixed dose combination [FDC]) administered once daily in human immunodeficiency virus (HIV) 1 infected adult participants that have not previously received antiretroviral therapy. The study is designed to demonstrate the non-inferior antiviral activity of DTG plus 3TC regimen to that of DTG plus TDF/FTC FDC and will characterise the long term antiviral activity, tolerability and safety of DTG plus 3TC through Week 148. Approximately, 700 participants will be randomised 1:1 to receive DTG + 3TC or DTG + TDF/FTC FDC. Participants will be stratified by screening HIV 1 ribonucleotide nucleic acid (RNA) levels and by screening CD4+ (cluster of differentiation 4) cell count.

ELIGIBILITY:
Inclusion Criteria:

* Must be an HIV 1 infected adult >=18 years of age (or older, if required by local regulations) at the time of signing the informed consent
* An eligible female participant should not be pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at Screening and negative urine test at Baseline), not lactating, and at least one of the following conditions applies

  * Non reproductive premenopausal women are those that have undergone documented tubal ligation or documented hysteroscopic tubal occlusion procedure with follow up confirmation of bilateral tubal occlusion or documented bilateral oophorectomy or hysterectomy
  * Non reproductive premenopausal women are those with 12 months of spontaneous amenorrhea and >=45 years of age
  * Women with reproductive potential agree to follow one of the protocol-defined methods for avoiding pregnancy
* Should have screening plasma HIV 1 RNA levels of 1000 c/mL to <=100,000 c/mL. If an independent review of accumulated data from other clinical trials investigating the DTG plus 3TC dual regimen is supportive of the DTG plus 3TC treatment regimen, enrolment will be opened to participants with Screening plasma HIV 1 RNA of 1000 c/mL to <=500,000 c/mL
* Participants should be antiretroviral naïve (defined as <=10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV 1 infection). Participants who received HIV post exposure prophylaxis (PEP) or pre exposure prophylaxis (PrEP) in the past are allowed as long as the last PEP/PrEP dose was >1 year from HIV diagnosis or there is documented HIV seronegativity between the last prophylactic dose and the date of HIV diagnosis
* Participant or the participants legal representative capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and the protocol
* Participants enrolled in France: a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria

* Women who are breastfeeding or plan to become pregnant or breastfeed during the study
* Any evidence of an active centers for disease control and prevention (CDC) Stage 3 disease (CDC, 2014), except cutaneous Kaposi's sarcoma not requiring systemic therapy and historical or current CD4 cell counts less than 200 cells/mm^3
* Participants with severe hepatic impairment (Class C) as determined by Child Pugh classification
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones
* Evidence of hepatitis B virus (HBV) infection or HBV surface antibody (anti-HBs or HBsAb) based on:

Participants positive for HBV surface antigen (HBsAg) at screening will be excluded Participants negative for HBV core antibody (anti HBs) but positive for anti HBc (negative HBsAg status) and positive for HBV deoxyribose nucleic acid (DNA) will be excluded; however, participants positive for anti HBc (negative HBsAg status) and positive for anti HBs (past and/or current evidence) are immune to HBV and will not be excluded

* Anticipated need for any hepatitis B virus (HCV) therapy during the first 48 weeks of the study and for HCV therapy based on interferon or any drugs that have a potential for adverse drug:drug interactions with study treatment throughout the entire study period
* Untreated syphilis infection positive RPR at Screening without clear documentation of treatment. Participants who are at least 14 days post completed treatment are eligible
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; other localised malignancies require agreement between the investigator and the Study Medical Monitor for inclusion of the participant
* Participants who in the Investigator's judgment, poses a significant suicidality risk. Recent history of suicidal behaviour and/or suicidal ideation may be considered as evidence of serious suicide risk
* Treatment with an HIV 1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any of the following agents within 28 days of Screening:

  * Radiation therapy,
  * Cytotoxic chemotherapeutic agents,
  * Any systemic immune suppressant
* Treatment with any agent, except recognised ART as allowed above, with documented activity against HIV 1 in vitro within 28 days of first dose of study treatment
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study treatment
* Participants enrolled in France: the participant has participated in any study using an investigational drug during the previous 60 days or 5 half lives, or twice the duration of the biological effect of the experimental drug or vaccine, whichever is longer, prior to screening for the study or the participant will participate simultaneously in another clinical study
* Any evidence of pre existing viral resistance based on the presence of any major resistance associated mutation in the Screening result or, if known, in any historical resistance test result
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening period to verify a result
* Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the participants participation in the study of an investigational compound
* Alanine aminotransferase (ALT) >=5 times the upper limit of normal (ULN) or ALT >=3xULN and bilirubin >=1.5xULN (with >35% direct bilirubin)
* Creatinine clearance of <50 mL/min per 1.73 m^2 via the chronic kidney disease epidemiology collaboration (CKD EPI) method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (77):
- United States (15):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Bellaire, Texas
- Argentina (3):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Australia (3):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Fortitude Valley, Queensland
- Belgium (2):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (4):
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (5):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (10):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Busto Arsizio (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Reggio Emilia
  - GSK Investigational Site, Roma
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Distrito Federal
- GSK Investigational Site, Rotterdam, Netherlands
- Portugal (3):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Romania (2):
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Galati
- Russia (6):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Toliyatti
  - GSK Investigational Site, Yekaterinburg
  - GSK Investigational Site, Красноярск
- GSK Investigational Site, Observatory, Cape Town, South Africa
- South Korea (3):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo
- Taiwan (2):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

REFERENCES:
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Derived] Ait-Khaled M, Sierra Madero J, Estrada V, Gulminetti R, Hagins D, Tsai HC, Man C, Sievers J, Grove R, Zolopa A, Wynne B, van Wyk J. Impact of treatment adherence on efficacy of dolutegravir plus lamivudine and dolutegravir plus tenofovir disoproxil fumarate/emtricitabine: pooled analysis of the GEMINI-1 and GEMINI-2 clinical studies. HIV Res Clin Pract. 2021 Dec 9;23(1):9-14. Epub 2021 Dec 16. PMID 34913844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a randomized, double-blind, parallel-group, non-inferiority study. The study consisted of double blind, open label, and continuation phase.
Pre-assignment Details: Total of 719 participants were enrolled and randomized. Five participants were randomized but not treated. A total of 714 participants received at least one dose of study treatment, following randomization creating the intent to treat exposed (ITT-E) population.
Groups:
- DTG + 3TC-Double Blind Phase: Participants received a two-drug regimen of dolutegravir plus lamivudine (DTG + 3TC) once daily for 96 weeks in the double blind phase
- DTG + TDF/FTC-Double Blind Phase: Participants received a three-drug regimen of dolutegravir plus tenofovir/emtricitabine (DTG + TDF/FTC) fixed dose combination (FDC) once daily for 96 weeks in the double blind phase.
- DTG + 3TC - Open-label Phase: Participants received a two-drug regimen of DTG + 3TC administered orally, once daily from Week 96 to Week 148 in the open-label phase.
- DTG + TDF/FTC - Open-label Phase: Participants received a three-drug regimen of DTG + TDF/FTC FDC administered orally, once daily from Week 96 to Week 148 in the open-label phase.
- DTG + 3TC - Continuation Phase: Participants received a DTG + 3TC administered orally, once daily from Week 148 to Week 280 in a continuation phase.
Period: Double-blind (Day 1 to Week 96)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase | DTG + 3TC - Open-label Phase | DTG + TDF/FTC - Open-label Phase | DTG + 3TC - Continuation Phase
Started (Randomized) | 359 | 360 | 0 | 0 | 0
Intent to Treat Exposed | 356 | 358 | 0 | 0 | 0
Completed | 301 | 320 | 0 | 0 | 0
Not Completed | 58 | 40 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 7 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 2 | 0 | 0 | 0
Not completed — Protocol Deviation | 6 | 6 | 0 | 0 | 0
Not completed — Protocol Withdrawal Criterion Met | 2 | 6 | 0 | 0 | 0
Not completed — Lost to Follow-up | 13 | 7 | 0 | 0 | 0
Not completed — Physician Decision | 9 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 6 | 0 | 0 | 0
Not completed — Randomized but not treated | 3 | 2 | 0 | 0 | 0
Period: Open-label Phase (Week 96 to Week 148)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase | DTG + 3TC - Open-label Phase | DTG + TDF/FTC - Open-label Phase | DTG + 3TC - Continuation Phase
Started | 0 | 0 | 301 | 319 (One participant who withdrew right after completion of double blind not 'Entered' open label phase.) | 0
Completed | 0 | 0 | 281 | 294 | 0
Not Completed | 0 | 0 | 20 | 25 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 6 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 0 | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 7 | 6 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 5 | 0
Period: Continuation Phase(Week 148 to Week 280)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase | DTG + 3TC - Open-label Phase | DTG + TDF/FTC - Open-label Phase | DTG + 3TC - Continuation Phase
Started | 0 | 0 | 0 | 0 | 233 (233 participants from the Open-label Phase entered in the Continuation Phase)
Completed | 0 | 0 | 0 | 0 | 212
Not Completed | 0 | 0 | 0 | 0 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 10
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for the Intent-to-Treat Exposed (ITT-E) Population which consisted of all randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase | Total
Number analyzed (Participants) | 356 | 358 | 714
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (9.88) | 35.0 (10.72) | 34.5 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 52 | 111
  Male | 297 | 306 | 603
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American (Am) Indian or Alaska (Al.) native | 31 | 28 | 59
  Race: Asian-Central/South Asian heritage (H.) | 0 | 4 | 4
  Race: Asian - East Asian H. | 33 | 36 | 69
  Race: Asian - South East Asian H. | 4 | 2 | 6
  Race: Black or African Am | 39 | 36 | 75
  Race: Native Hawaiian or other Pacific Islander | 2 | 0 | 2
  Race: White (Wt)-Arabic/North African H. | 5 | 5 | 10
  Race: White - White/Caucasian/European H. | 239 | 242 | 481
  Race: Multiple | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/mL (c/mL) at Week 48
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using Food and Drug Administration (FDA) Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant antiretroviral therapy (ART) prior to the visit of interest. This endpoint was analyzed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights. Intent-To-Treat Exposed (ITT-E) Population was used which comprised of all randomized participants who received at least one dose of study treatment. Percentage values are rounded to the nearest whole digit.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants | 90 [86.8 to 93.0] | 93 [90.0 to 95.4]
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Non-Inferiority — Treatment with DTG+ 3TC was to be declared non-inferior to treatment with DTG+TDF/FTC if the lower end of a two-sided 95% confidence interval for the difference between the two groups in response rates at Week 48 greater than -10%; Adjusted difference in proportion = -2.6, 95% CI 2-sided [-6.7 to 1.5] — Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<=versus [vs.]>100,000 c/mL) and cluster of differentiation 4+ (CD4+) cell count (<= vs. >200 cells per cubic millimeter)

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 24
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. This endpoint was analyzed using a stratified analysis with Cochran-Mantel-Haenszel weights. Percentage values are rounded to the nearest whole digit.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants | 92 [89.7 to 95.2] | 93 [90.4 to 95.7]
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Adjusted difference in proportion = -0.4, 95% CI 2-sided [-4.2 to 3.4] — Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<=vs.>100,000 c/mL) and CD4+ cell count (<= vs. >200 cells per cubic millimeter)

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 96
Description: as for outcome 2
Time Frame: Week 96
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- DTG + 3TC-Double Blind Phase: Participants received a two-drug regimen of dolutegravir plus lamivudine (DTG + 3TC) once daily for 96 weeks in double blind phase
- DTG + TDF/FTC-Double Blind Phase: Participants received a three-drug regimen of dolutegravir plus tenofovir/emtricitabine (DTG + TDF/FTC) fixed dose combination (FDC) once daily for 96 weeks in double blind phase.
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants | 84 [80.5 to 88.1] | 89 [86.2 to 92.6]
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Adjusted difference in proportion = -4.9, 95% CI 2-sided [-9.8 to 0.0] — Week 96. Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<= vs. >100,000 c/mL) and CD4+ cell count (<= vs. >200 cells/mm^3)

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 144
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. This endpoint was analyzed using a stratified analysis with CMH weights. Percentage values are rounded to the nearest whole digit.
Time Frame: Week 144
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- DTG + 3TC - Double-blind Phase + Open-label Phase: Participants received a two-drug regimen of DTG + 3TC administered orally, once daily until Week 96 in double-blind phase and participants continued to receive DTG + 3TC from Week 96 to Week 148 in an open-label phase.
- DTG + TDF/FTC - Double-blind Phase + Open-label Phase: Participants received a three-drug regimen of DTG + TDF/FTC FDC administered orally, once daily until Week 96 in double-blind phase and participants continued to receive DTG + TDF/FTC FDC from Week 96 to Week 148 in an open-label phase.
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants | 79 [74.7 to 83.2] | 83 [78.8 to 86.6]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Adjusted difference in proportion = -3.6, 95% CI 2-sided [-9.4 to 2.1] — Week 144. Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<= vs. >100,000 c/mL) and CD4+ cell count (<= vs. >200 cells/mm^3)

5. Secondary Outcome: Time to Viral Suppression (HIV-1 RNA <50 c/mL) up to Week 144
Description: Time of viral suppression is defined as the first viral load value <50 c/mL. Nonparametric Kaplan-Meier method was performed. Participants who withdrew for any reason without being suppressed were censored at date of withdrawal. Participants who have not been withdrawn and have not had viral suppression at time of the analysis were censored at last viral load date. Confidence Interval (CI) was estimated using the Brookmeyer-Crowley method.
Time Frame: Up to Week 144
Population: ITT-E Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Days | 29.0 [29.0 to 53.0] | 29.0 [29.0 to 56.0]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.658, Generalized Wilcoxon procedure — The generalized Wilcoxon procedure was used to estimate a p-value for detecting a difference in cumulative incidence curves between treatment groups; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.86 to 1.16] — Hazard ratios were estimated using the Cox proportional hazard regression model

6. Secondary Outcome: CD4+ Cell Counts at Weeks 24 and 48
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry.
Time Frame: Weeks 24 and 48
Population: ITT-E Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter (cells/mm^3)
Groups:
- DTG + 3TC Double Blind Phase: Participants received a two-drug regimen of dolutegravir plus lamivudine (DTG + 3TC) once daily for 96 weeks in double blind phase
Arm/Group | DTG + 3TC Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Cells per cubic millimeter (cells/mm^3)
  Week 24, n=340,341: number analyzed (Participants) | 340 | 341
  Week 24, n=340,341 | 655.3 (288.32) | 632.8 (262.61)
  Week 48, n=324,334: number analyzed (Participants) | 324 | 334
  Week 48, n=324,334 | 687.7 (275.47) | 675.3 (274.46)

7. Secondary Outcome: CD4+ Cell Counts at Week 96
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+ cells. Analysis was performed by flow cytometry.
Time Frame: Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter (cells/mm^3)
Groups:
- DTG + 3TC Double Blind Phase: Participants received a two-drug regimen of dolutegravir plus lamivudine (DTG + 3TC) once daily for 96 weeks in the double blind phase
Arm/Group | DTG + 3TC Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 301 | 320
Cells per cubic millimeter (cells/mm^3) | 732.8 (298.05) | 711.5 (284.15)

8. Secondary Outcome: CD4+ Cell Counts at Week 144
Description: as for outcome 7
Time Frame: Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 270 | 287
Cells per cubic millimeter (cells/mm^3) | 767.8 (274.00) | 758.2 (285.35)

9. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 24 and 48
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is defined as the the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error has been presented. Adjusted mean is the estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for the following covariates/factors: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction, and Baseline CD4+ cell count and visit interaction, with visit as the repeated factor.
Time Frame: Baseline (Day 1) and Weeks 24, 48
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells per cubic millimeter
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Cells per cubic millimeter
  Week 24, n=340,341: number analyzed (Participants) | 340 | 341
  Week 24, n=340,341 | 192.2 (9.67) | 175.1 (9.41)
  Week 48, n=324,334: number analyzed (Participants) | 324 | 334
  Week 48, n=324,334 | 222.2 (9.87) | 217.7 (10.64)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.206, Mixed Model Repeated Measures (MMRM); Mean Difference (Net) = 17.1, 95% CI 2-sided [-9.4 to 43.6] — Week 24. Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.754, Mixed Model Repeated Measures (MMRM); Mean Difference (Net) = 4.6, 95% CI 2-sided [-23.9 to 33.0] — Week 48. Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor

10. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 96
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+ cells. Analysis was performed by flow cytometry. Baseline value is defined as the the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error has been presented. Adjusted mean is the estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for the following covariates/factors: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction, and Baseline CD4+ cell count and visit interaction, with visit as the repeated factor.
Time Frame: Baseline (Day 1) and Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Cells per cubic millimeter
Groups:
- DTG + 3TC - Double-blind Phase: Participants received a two-drug regimen of dolutegravir plus lamivudine (DTG + 3TC) once daily for 96 weeks in the double blind phase
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 301 | 320
Cells per cubic millimeter | 264.7 (11.32) | 253.8 (11.40)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.500, Mixed Model Repeated Measures (MMRM); Mean Difference (Net) = 10.8, 95% CI 2-sided [-20.7 to 42.4] — Week 96. Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor

11. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 144
Description: as for outcome 10
Time Frame: Baseline (Day 1) and Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Cells per cubic millimeter
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 270 | 287
Cells per cubic millimeter | 301.8 (11.51) | 303.2 (12.13)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.934, Mixed Model Repeated Measures (MMRM); Mean Difference (Net) = -1.4, 95% CI 2-sided [-34.2 to 31.5] — Week 144.Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor

12. Secondary Outcome: Number of Participants With HIV-1 Disease Progression up to Week 144
Description: HIV-associated conditions were recorded during the study and was assessed according to the 2014 Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection in Adults. Disease progressions summarize participants who had HIV infection stage 3 associated conditions or death. Indicators of clinical disease progression were defined as: CDC Category Stage 1 at enrollment to Stage 3 event; CDC Category Stage 2 at enrolment to Stage 3 event; CDC Category Stage 3 at enrollment to New Stage 3 Event; CDC Category Stage 1, 2 or 3 at enrolment to Death.
Time Frame: Up to Week 144
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Participants
  No HIV-1 disease progression | 352 | 356
  From CDC Stage 1 to CDC Stage 3 Event | 0 | 0
  From CDC Stage 2 to CDC Stage 3 Event | 2 | 2
  From CDC Stage 3 to New CDC Stage 3 Event | 1 | 0
  From CDC Stage 1, 2 or 3 to Death | 1 | 0

13. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance up to Week 144
Description: Number of participants, who met confirmed virologic withdrawal (CVW) criteria, with treatment emergent genotypic resistance to Integrase strand transfer inhibitor (INSTI) and/or Nucleoside reverse transcriptase inhibitor (NRTI) was summarized. The Viral Genotypic Population comprised of all participants in the ITT-E population who have available on-treatment genotypic resistance data.
Time Frame: Up to Week 144
Population: Viral Genotypic Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 8 | 8
Participants
  INSTI Mutations | 0 | 0
  Major mutations of NRTI | 0 | 0

14. Secondary Outcome: Number of Participants With Treatment-emergent Phenotypic Resistance up to Week 144
Description: Number of participants, who meet CVW criteria, with treatment emergent phenotypic resistance to INSTI and/or NRTI were summarized. Assessment of antiviral activity of anti-retroviral therapy (ART) using phenotypic test results was interpreted through a proprietary algorithm (from Monogram Biosciences) and provides the overall susceptibility of the drug. Partially sensitive and resistant calls were considered resistant in this analysis. The Viral Phenotypic Population comprised of all participants in the ITT-E population who have available on-treatment phenotypic resistance data.
Time Frame: Up to Week 144
Population: Viral Phenotypic Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 5 | 6
Participants
  INSTI, DTG, Sensitive, n=,5,4: number analyzed (Participants) | 5 | 4
  INSTI, DTG, Sensitive, n=,5,4 | 5 | 4
  INSTI, DTG, Resistant, n=5,4: number analyzed (Participants) | 5 | 4
  INSTI, DTG, Resistant, n=5,4 | 0 | 0
  INSTI, EGV, Sensitive, n=5,4: number analyzed (Participants) | 5 | 4
  INSTI, EGV, Sensitive, n=5,4 | 5 | 4
  INSTI, EGV, Resistant, n=5,4: number analyzed (Participants) | 5 | 4
  INSTI, EGV, Resistant, n=5,4 | 0 | 0
  INSTI, RAL, Sensitive, n=5,4: number analyzed (Participants) | 5 | 4
  INSTI, RAL, Sensitive, n=5,4 | 5 | 4
  INSTI, RAL, Resistant, n=5,4: number analyzed (Participants) | 5 | 4
  INSTI, RAL, Resistant, n=5,4 | 0 | 0
  NRTI, 3TC, Sensitive, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, 3TC, Sensitive, n=5,5 | 5 | 5
  NRTI, 3TC, Resistant, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, 3TC, Resistant, n=5,5 | 0 | 0
  NRTI, ABC, Sensitive, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, ABC, Sensitive, n=5,5 | 5 | 5
  NRTI, ABC, Resistant, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, ABC, Resistant, n=5,5 | 0 | 0
  NRTI, AZT, Sensitive, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, AZT, Sensitive, n=5,5 | 5 | 5
  NRTI, AZT, Resistant, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, AZT, Resistant, n=5,5 | 0 | 0
  NRTI, D4T, Sensitive, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, D4T, Sensitive, n=5,5 | 5 | 5
  NRTI, D4T, Resistant, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, D4T, Resistant, n=5,5 | 0 | 0
  NRTI, DDI, Sensitive, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, DDI, Sensitive, n=5,5 | 5 | 5
  NRTI, DDI, Resistant, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, DDI, Resistant, n=5,5 | 0 | 0
  NRTI, FTC, Sensitive, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, FTC, Sensitive, n=5,5 | 5 | 5
  NRTI, FTC, Resistant, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, FTC, Resistant, n=5,5 | 0 | 0
  NRTI, TDF, Sensitive, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, TDF, Sensitive, n=5,5 | 5 | 5
  NRTI, TDF, Resistant, n=5,5: number analyzed (Participants) | 5 | 5
  NRTI, TDF, Resistant, n=5,5 | 0 | 0

15. Secondary Outcome: Number of Participants With Any AE and SAE up to Week 148
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or protocol defined event associated with liver injury and impaired liver function were categorized as SAE. Safety Population was used which comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Week 148
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Participants
  Any AE | 307 | 316
  Any SAE | 37 | 38

16. Secondary Outcome: Number of Participants With AEs by Maximum Severity Grades up to Week 144
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were evaluated by the investigator and graded according to the DAIDS toxicity scales from Grade 1 to 5 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms. Number of participants with adverse events by maximum grade have been presented.
Time Frame: Up to Week 144
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Participants
  Grade 1 AEs | 33 | 35
  Grade 2 AEs | 229 | 242
  Grade 3 AEs | 37 | 34
  Grade 4 AEs | 7 | 5
  Grade 5 AEs | 1 | 0

17. Secondary Outcome: Number of Participants With Any Drug Related AEs and Drug Related AEs by Maximum Grade up to Week 144
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were evaluated by the investigator and graded according to the DAIDS toxicity scales from Grade 1 to 5. (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms. Number of participants with drug related AEs and drug related AEs by by maximum grade have been presented.
Time Frame: Up to Week 144
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Participants
  Any drug related AE | 77 | 101
  Drug related AEs with maximum toxicity Grade 1 | 51 | 70
  Drug related AEs with maximum toxicity Grade 2 | 19 | 28
  Drug related AEs with maximum toxicity Grade 3 | 7 | 3
  Drug related AEs with maximum toxicity Grade 4 | 0 | 0
  Drug related AEs with maximum toxicity Grade 5 | 0 | 0

18. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities up to Week 144
Description: Blood samples were collected up to Week 144 for assessment of hemoglobin, leukocytes, neutrophils and platelets. Any abnormality was graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Only those participants with maximum post-Baseline emergent hematology toxicities in any of the listed hematology parameters have been presented.
Time Frame: Up to Week 144
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Participants
  Hemoglobin, Grades 1 to 4 | 9 | 7
  Hemoglobin, Grades 2 to 4 | 1 | 1
  Hemoglobin, Grades 3 to 4 | 0 | 0
  Hemoglobin, Grade 1 | 8 | 6
  Hemoglobin, Grade 2 | 1 | 1
  Hemoglobin, Grade 3 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0
  Leukocytes, Grades 1 to 4 | 16 | 3
  Leukocytes, Grades 2 to 4 | 4 | 2
  Leukocytes, Grades 3 to 4 | 0 | 0
  Leukocytes, Grade 1 | 12 | 1
  Leukocytes, Grade 2 | 4 | 2
  Leukocytes, Grade 3 | 0 | 0
  Leukocytes, Grade 4 | 0 | 0
  Neutrophils, Grades 1 to 4 | 25 | 18
  Neutrophils, Grades 2 to 4 | 19 | 11
  Neutrophils, Grades 3 to 4 | 7 | 6
  Neutrophils, Grade 1 | 6 | 7
  Neutrophils, Grade 2 | 12 | 5
  Neutrophils, Grade 3 | 5 | 5
  Neutrophils, Grade 4 | 2 | 1
  Platelets, Grades 1 to 4 | 14 | 11
  Platelets, Grades 2 to 4 | 8 | 4
  Platelets, Grades 3 to 4 | 1 | 1
  Platelets, Grade 1 | 6 | 7
  Platelets, Grade 2 | 7 | 3
  Platelets, Grade 3 | 0 | 1
  Platelets, Grade 4 | 1 | 0

19. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Chemistry Toxicities up to Week 144
Description: Blood samples were collected up to Week 144 for assessment of Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase (ALP), Aspartate aminotransferase (AST), Bilirubin, Carbon dioxide (CO2), Cholesterol, Creatine kinase (CK), Creatinine, Direct Bilirubin, Glomerular filtration rate (GFR) from creatinine adjusted for body surface area (BSA), Hypercalcemia, Hyperglycemia, Hyperkalemia, Hypernatremia, Hypocalcemia, Hypoglycemia, Hypokalemia, Hyponatremia, Low density lipid (LDL) Cholesterol, Lactate Dehydrogenase, Lipase, Phosphate, and Triglycerides. Any abnormality was graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Only those participants with maximum post-Baseline emergent chemistry toxicities in any of the chemistry parameters have been presented
Time Frame: Up to Week 144
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Participants
  ALT, Grades 1 to 4 | 55 | 81
  ALT, Grades 2 to 4 | 23 | 25
  ALT, Grades 3 to 4 | 14 | 9
  ALT, Grade 1 | 32 | 56
  ALT, Grade 2 | 9 | 16
  ALT, Grade 3 | 7 | 4
  ALT, Grade 4 | 7 | 5
  Albumin, Grades 1 to 4 | 1 | 1
  Albumin, Grades 2 to 4 | 1 | 0
  Albumin, Grades 3 to 4 | 0 | 0
  Albumin, Grade 1 | 0 | 1
  Albumin, Grade 2 | 1 | 0
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  ALP, Grades 1 to 4 | 8 | 10
  ALP, Grades 2 to 4 | 3 | 1
  ALP, Grades 3 to 4 | 0 | 0
  ALP, Grade 1 | 5 | 9
  ALP, Grade 2 | 3 | 1
  ALP, Grade 3 | 0 | 0
  ALP, Grade 4 | 0 | 0
  AST, Grades 1 to 4 | 52 | 79
  AST, Grades 2 to 4 | 27 | 31
  AST, Grades 3 to 4 | 8 | 13
  AST, Grade 1 | 25 | 48
  AST, Grade 2 | 19 | 18
  AST, Grade 3 | 6 | 9
  AST, Grade 4 | 2 | 4
  Bilirubin, Grades 1 to 4 | 42 | 51
  Bilirubin, Grades 2 to 4 | 14 | 17
  Bilirubin, Grades 3 to 4 | 4 | 4
  Bilirubin, Grade 1 | 28 | 34
  Bilirubin, Grade 2 | 10 | 13
  Bilirubin, Grade 3 | 2 | 4
  Bilirubin, Grade 4 | 2 | 0
  CO2, Grades 1 to 4 | 126 | 116
  CO2, Grades 2 to 4 | 8 | 9
  CO2, Grades 3 to 4 | 0 | 0
  CO2, Grade 1 | 118 | 107
  CO2, Grade 2 | 8 | 9
  CO2, Grade 3 | 0 | 0
  CO2, Grade 4 | 0 | 0
  Cholesterol, Grades 1 to 4 | 77 | 40
  Cholesterol, Grades 2 to 4 | 24 | 13
  Cholesterol, Grades 3 to 4 | 0 | 1
  Cholesterol, Grade 1 | 53 | 27
  Cholesterol, Grade 2 | 24 | 12
  Cholesterol, Grade 3 | 0 | 1
  Cholesterol, Grade 4 | 0 | 0
  CK, Grades 1 to 4 | 76 | 75
  CK, Grades 2 to 4 | 43 | 52
  CK, Grades 3 to 4 | 26 | 36
  CK, Grade 1 | 33 | 23
  CK, Grade 2 | 17 | 16
  CK, Grade 3 | 15 | 21
  CK, Grade 4 | 11 | 15
  Creatinine, Grades 1 to 4 | 21 | 31
  Creatinine, Grades 2 to 4 | 1 | 3
  Creatinine, Grades 3 to 4 | 0 | 2
  Creatinine, Grade 1 | 20 | 28
  Creatinine, Grade 2 | 1 | 1
  Creatinine, Grade 3 | 0 | 2
  Creatinine, Grade 4 | 0 | 0
  Direct Bilirubin, Grades 1 to 4 | 14 | 13
  Direct Bilirubin, Grades 2 to 4 | 14 | 13
  Direct Bilirubin, Grades 3 to 4 | 14 | 13
  Direct Bilirubin, Grade 1 | 0 | 0
  Direct Bilirubin, Grade 2 | 0 | 0
  Direct Bilirubin, Grade 3 | 14 | 13
  Direct Bilirubin, Grade 4 | 0 | 0
  GFR from creatinine adjusted for BSA Grades 1 to 4 | 185 | 226
  GFR from creatinine adjusted for BSA Grades 2 to 4 | 185 | 226
  GFR from creatinine adjusted for BSA Grades 3 to 4 | 13 | 27
  GFR from creatinine adjusted for BSA, Grade 1 | 0 | 0
  GFR from creatinine adjusted for BSA, Grade 2 | 172 | 199
  GFR from creatinine adjusted for BSA Grades 3 | 13 | 25
  GFR from creatinine adjusted for BSA, Grade 4 | 0 | 2
  Hypercalcaemia, Grades 1 to 4 | 7 | 4
  Hypercalcaemia, Grades 2 to 4 | 0 | 0
  Hypercalcaemia, Grades 3 to 4 | 0 | 0
  Hypercalcaemia, Grade 1 | 7 | 4
  Hypercalcaemia, Grade 2 | 0 | 0
  Hypercalcaemia, Grade 3 | 0 | 0
  Hypercalcaemia, Grade 4 | 0 | 0
  Hyperglycemia, Grades 1 to 4 | 91 | 81
  Hyperglycemia, Grades 2 to 4 | 38 | 25
  Hyperglycemia, Grades 3 to 4 | 3 | 2
  Hyperglycemia, Grade 1 | 53 | 56
  Hyperglycemia, Grade 2 | 35 | 23
  Hyperglycemia, Grade 3 | 3 | 2
  Hyperglycemia, Grade 4 | 0 | 0
  Hyperkalemia, Grades 1 to 4 | 1 | 4
  Hyperkalemia, Grades 2 to 4 | 0 | 1
  Hyperkalemia, Grades 3 to 4 | 0 | 1
  Hyperkalemia, Grade 1 | 1 | 3
  Hyperkalemia, Grade 2 | 0 | 0
  Hyperkalemia, Grade 3 | 0 | 0
  Hyperkalemia, Grade 4 | 0 | 1
  Hypernatremia, Grades 1 to 4 | 6 | 3
  Hypernatremia, Grades 2 to 4 | 0 | 0
  Hypernatremia, Grades 3 to 4 | 0 | 0
  Hypernatremia, Grade 1 | 6 | 3
  Hypernatremia, Grade 2 | 0 | 0
  Hypernatremia, Grade 3 | 0 | 0
  Hypernatremia, Grade 4 | 0 | 0
  Hypocalcaemia, Grades 1 to 4 | 14 | 13
  Hypocalcaemia, Grades 2 to 4 | 4 | 3
  Hypocalcaemia, Grades 3 to 4 | 0 | 1
  Hypocalcaemia, Grade 1 | 10 | 10
  Hypocalcaemia, Grade 2 | 4 | 2
  Hypocalcaemia, Grade 3 | 0 | 1
  Hypocalcaemia, Grade 4 | 0 | 0
  Hypoglycemia, Grades 1 to 4 | 22 | 17
  Hypoglycemia, Grades 2 to 4 | 8 | 3
  Hypoglycemia, Grades 3 to 4 | 2 | 1
  Hypoglycemia, Grade 1 | 14 | 14
  Hypoglycemia, Grade 2 | 6 | 2
  Hypoglycemia, Grade 3 | 1 | 0
  Hypoglycemia, Grade 4 | 1 | 1
  Hypokalemia, Grades 1 to 4 | 6 | 7
  Hypokalemia, Grades 2 to 4 | 0 | 1
  Hypokalemia, Grades 3 to 4 | 0 | 0
  Hypokalemia, Grade 1 | 6 | 6
  Hypokalemia, Grade 2 | 0 | 1
  Hypokalemia, Grade 3 | 0 | 0
  Hypokalemia, Grade 4 | 0 | 0
  Hyponatremia, Grades 1 to 4 | 25 | 28
  Hyponatremia, Grades 2 to 4 | 2 | 0
  Hyponatremia, Grades 3 to 4 | 0 | 0
  Hyponatremia, Grade 1 | 23 | 28
  Hyponatremia, Grade 2 | 2 | 0
  Hyponatremia, Grade 3 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 0
  LDL Cholesterol, Grades 1 to 4 | 57 | 35
  LDL Cholesterol, Grades 2 to 4 | 17 | 14
  LDL Cholesterol, Grades 3 to 4 | 5 | 4
  LDL Cholesterol, Grade 1 | 40 | 21
  LDL Cholesterol, Grade 2 | 12 | 10
  LDL Cholesterol, Grade 3 | 5 | 4
  LDL Cholesterol, Grade 4 | 0 | 0
  Lactate Dehydrogenase, Grades 1 to 4 | 3 | 5
  Lactate Dehydrogenase, Grades 2 to 4 | 0 | 1
  Lactate Dehydrogenase, Grades 3 to 4 | 0 | 0
  Lactate Dehydrogenase, Grade 1 | 3 | 4
  Lactate Dehydrogenase, Grade 2 | 0 | 1
  Lactate Dehydrogenase, Grade 3 | 0 | 0
  Lactate Dehydrogenase, Grade 4 | 0 | 0
  Lipase, Grades 1 to 4 | 65 | 80
  Lipase, Grades 2 to 4 | 35 | 49
  Lipase, Grades 3 to 4 | 10 | 18
  Lipase, Grade 1 | 30 | 31
  Lipase, Grade 2 | 25 | 31
  Lipase, Grade 3 | 8 | 10
  Lipase, Grade 4 | 2 | 8
  Phosphate, Grades 1 to 4 | 70 | 68
  Phosphate, Grades 2 to 4 | 35 | 47
  Phosphate, Grades 3 to 4 | 2 | 6
  Phosphate, Grade 1 | 35 | 21
  Phosphate, Grade 2 | 33 | 41
  Phosphate, Grade 3 | 2 | 6
  Phosphate, Grade 4 | 0 | 0
  Triglycerides, Grades 1 to 4 | 80 | 62
  Triglycerides, Grades 2 to 4 | 12 | 14
  Triglycerides, Grades 3 to 4 | 7 | 3
  Triglycerides, Grade 1 | 68 | 48
  Triglycerides, Grade 2 | 5 | 11
  Triglycerides, Grade 3 | 6 | 2
  Triglycerides, Grade 4 | 1 | 1

20. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to AEs Over Weeks 24, 48, 96
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. . Number of participants who discontinued treatment due to AEs have been reported.
Time Frame: Up to Week 24, Week 48 and Week 96
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Participants
  Up to Week 24 | 6 | 4
  Up to Week 48 | 7 | 8
  Up to Week 96 | 14 | 11

21. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to AEs Over Week 144
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants who discontinued treatment due to AEs have been reported.
Time Frame: Up to Week 144
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Participants | 18 | 17

22. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum Cystatin C and Serum Retinol Binding Protein (RBP) at Weeks 24, 48
Description: Blood and/or urine were collected to perform evaluation of renal inflammation biomarkers which included Serum Cystatin C and Serum Retinol Binding Protein (RBP). Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, baseline plasma HIV-1 RNA (factor), baseline CD4+ cell count (factor), age, sex (factor), race (factor), presence of diabetes mellitus (factor), presence of hypertension (factor), baseline biomarker value, treatment and visit interaction, and baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Error); unit: Milligrams per Liter (mg/L)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Milligrams per Liter (mg/L)
  Serum Cystatin C, Week 24, n=338, 336: number analyzed (Participants) | 338 | 336
  Serum Cystatin C, Week 24, n=338, 336 | -0.05 (0.007) | -0.03 (0.007)
  Serum Cystatin C, Week 48, n=324, 332: number analyzed (Participants) | 324 | 332
  Serum Cystatin C, Week 48, n=324, 332 | -0.07 (0.007) | -0.04 (0.006)
  Serum RBP, Week 24, n=332, 334: number analyzed (Participants) | 332 | 334
  Serum RBP, Week 24, n=332, 334 | 1.6 (0.41) | 1.9 (0.51)
  Serum RBP, Week 48, n=322, 332: number analyzed (Participants) | 322 | 332
  Serum RBP, Week 48, n=322, 332 | 0.5 (0.47) | 0.6 (0.46)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.025, Mixed Model Repeated Measures; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.04 to 0.00] — Serum Cystatin C, Week 24
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.05 to -0.01] — Serum Cystatin C, Week 48
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.683, Mixed Model Repeated Measures; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.6 to 1.0] — Serum RBP, Week 24
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.930, Mixed Model Repeated Measures; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.4 to 1.2] — Serum RBP, Week 48

23. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum Cystatin C at Week 96
Description: Blood samples were collected to perform evaluation of renal inflammation biomarkers which included Serum Cystatin C . Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, baseline plasma HIV-1 RNA (factor), baseline CD4+ cell count (factor), age, sex (factor), race (factor), presence of diabetes mellitus (factor), presence of hypertension (factor), baseline biomarker value, treatment and visit interaction, and baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Milligrams per Liter (mg/L)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 300 | 319
Milligrams per Liter (mg/L) | -0.11 (0.006) | -0.09 (0.006)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.009, Mixed Model Repeated Measures; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.04 to -0.01] — Week 96. Serum Cystatin C

24. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum Cystatin C at Week 144
Description: Blood samples were collected to perform evaluation of renal biomarkers which included Serum Cystatin C. Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Milligrams per Liter (mg/L)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 283 | 298
Milligrams per Liter (mg/L) | -0.12 (0.006) | -0.11 (0.007)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.108, Mixed Model Repeated Measures; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to -0.00] — Week 144. Serum Cystatin C

25. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum RBP at Week 96
Description: Blood and/or urine samples were collected to perform evaluation of renal biomarkers which included Serum RBP. Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per millimoles (ug/mmol)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 288 | 310
Microgram per millimoles (ug/mmol) | 1.535 (8.5872) | 7.704 (41.9650)

26. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum RBP at Week 144
Description: as for outcome 25
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per millimoles (ug/mmol)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 276 | 292
Microgram per millimoles (ug/mmol) | 1.760 (5.7909) | 8.855 (35.5147)

27. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum GFR From Cystatin C Adjusted Using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) and Serum or Plasma GFR From Creatinine Adjusted Using CKD-EPI at Weeks 24, 48
Description: Blood and/or urine were collected to perform evaluation of renal inflammation biomarkers which included Serum GFR from cystatin C adjusted using CKD-EPI (GFR-cystatin C adjusted)and Serum or Plasma GFR from creatinine adjusted using CKD-EPI. Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, baseline plasma HIV-1 RNA (factor), baseline CD4+ cell count (factor), age, sex (factor), race (factor), presence of diabetes mellitus (factor), presence of hypertension (factor), baseline biomarker value, treatment and visit interaction, and baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Milliliter/minute/1.73*meter^2
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Milliliter/minute/1.73*meter^2
  GFR-cystatin C adjusted, Week 24, n=338, 336: number analyzed (Participants) | 338 | 336
  GFR-cystatin C adjusted, Week 24, n=338, 336 | 4.4 (0.63) | 2.2 (0.60)
  GFR-cystatin C adjusted, Week 48, n=324, 332: number analyzed (Participants) | 324 | 332
  GFR-cystatin C adjusted, Week 48, n=324, 332 | 7.0 (0.60) | 4.1 (0.59)
  GFR-creatinine adjusted, Week 24, n=340, 341: number analyzed (Participants) | 340 | 341
  GFR-creatinine adjusted, Week 24, n=340, 341 | -13.5 (0.59) | -16.7 (0.56)
  GFR-creatinine adjusted, Week 48, n=326,335: number analyzed (Participants) | 326 | 335
  GFR-creatinine adjusted, Week 48, n=326,335 | -12.1 (0.56) | -15.6 (0.55)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.011, Mixed Model Repeated Measures; Mean Difference (Net) = 2.2, 95% CI 2-sided [0.5 to 4.0] — GFR-cystatin C adjusted, Week 24
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = 2.8, 95% CI 2-sided [1.2 to 4.5] — GFR-cystatin C adjusted, Week 48
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = 3.2, 95% CI 2-sided [1.6 to 4.8] — GFR-creatinine adjusted, Week 24
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = 3.5, 95% CI 2-sided [2.0 to 5.1] — GFR- creatinine adjusted, Week 48

28. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum GFR From Cystatin C Adjusted Using CKD-EPI and Serum or Plasma GFR From Creatinine Adjusted for BSA Using CKD-EPI Method at Week 96
Description: Blood samples were collected to perform evaluation of renal biomarkers which included Serum GFR from cystatin C adjusted using CKD-EPI and Serum or Plasma GFR from creatinine adjusted for BSA using CKD-EPI. Baseline value is the latest pre-dose Assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter/minute/1.73*meter^2
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 300 | 319
Milliliter/minute/1.73*meter^2
  GFR Cystatin C adjusted, Week 96 | 11.3 (14.54) | 9.3 (13.78)
  GFR creatinine adjusted, Week 96 | -15.3 (11.50) | -19.0 (11.25)

29. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum GFR From Cystatin C Adjusted Using CKD-EPI and Serum or Plasma GFR From Creatinine Adjusted for BSA Using CKD-EPI Method at Week 144
Description: as for outcome 28
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter/minute/1.73*meter^2
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Milliliter/minute/1.73*meter^2
  GFR Cystatin C adjusted, Week 144, n=283,298: number analyzed (Participants) | 283 | 298
  GFR Cystatin C adjusted, Week 144, n=283,298 | 13.0 (13.64) | 12.1 (15.24)
  GFR creatinine adjusted, Week 144, n=271, 289: number analyzed (Participants) | 271 | 289
  GFR creatinine adjusted, Week 144, n=271, 289 | -16.7 (11.65) | -19.3 (11.07)

30. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum or Plasma Creatinine at Weeks 24, 48
Description: Blood and/or urine were collected to perform evaluation of renal inflammation biomarker which included Serum or Plasma Creatinine. Baseline value is defined as the latest pre-dose assessment (Day 1). Change from Baseline was calculated as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, baseline plasma HIV-1 RNA (factor), baseline CD4+ cell count (factor), age, sex (factor), race (factor), presence of diabetes mellitus (factor), presence of hypertension (factor), baseline biomarker value, treatment and visit interaction, and baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Micromoles per Liter (umol/L)
Groups:
- DTG + 3TC-Double Blind Phase: Participants received a two-drug regimen of dolutegravir plus lamivudine (DTG + 3TC) once daily for96 weeks in the double blind phase
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Micromoles per Liter (umol/L)
  Serum or Plasma Creatinine, Week 24, n=340, 343: number analyzed (Participants) | 340 | 343
  Serum or Plasma Creatinine, Week 24, n=340, 343 | 11.88 (0.510) | 15.07 (0.520)
  Serum or Plasma Creatinine, Week 48, n=326, 335: number analyzed (Participants) | 326 | 335
  Serum or Plasma Creatinine, Week 48, n=326, 335 | 10.39 (0.466) | 13.61 (0.480)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -3.19, 95% CI 2-sided [-4.62 to -1.75] — Week 24
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -3.22, 95% CI 2-sided [-4.54 to -1.91] — Week 48

31. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum or Plasma Creatinine at Week 96
Description: as for outcome 30
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Micromoles per Liter (umol/L)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 300 | 319
Micromoles per Liter (umol/L) | 12.75 (0.623) | 16.10 (0.539)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -3.34, 95% CI 2-sided [-4.96 to -1.72] — Week 96. Serum or Plasma creatinine

32. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum or Plasma Creatinine at Week 144
Description: as for outcome 30
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Micromoles per Liter (umol/L)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 271 | 289
Micromoles per Liter (umol/L) | 12.89 (0.583) | 15.87 (0.560)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -2.98, 95% CI 2-sided [-4.57 to -1.40] — Week 144. Serum or Plasma creatinine

33. Secondary Outcome: Ratio to Baseline in Renal Biomarkers-Urine and Serum Beta-2 Microglobulin (B2M), Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine, Urine RBP 4 and Urine RBP 4/Urine Creatinine at Weeks 24, 48
Description: Blood and/or urine were collected to perform evaluation of renal inflammation biomarkers which included Urine and Serum B2M, Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine, Urine RBP 4 and Urine RBP 4/Urine Creatinine. Baseline value is defined as the latest pre-dose assessment (Day 1). Ratio to Baseline was calculated as ratio of post-dose visit value over Baseline value. Statistical analysis of changes from baseline were performed on log-transformed data. Results were transformed back via exponential transformation such that treatment comparisons are assessed via odds ratios. Estimated ratio of geometric means (each visit over Baseline) and 95% confidence interval (CI) have been presented.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Ratio
  Serum B2M, Week 24, n=338, 335: number analyzed (Participants) | 338 | 335
  Serum B2M, Week 24, n=338, 335 | 0.798 [0.779 to 0.817] | 0.872 [0.856 to 0.890]
  Serum B2M, Week 48, n=324, 332: number analyzed (Participants) | 324 | 332
  Serum B2M, Week 48, n=324, 332 | 0.806 [0.790 to 0.823] | 0.892 [0.876 to 0.908]
  Urine B2M, Week 24, n=121, 95: number analyzed (Participants) | 121 | 95
  Urine B2M, Week 24, n=121, 95 | 0.887 [0.756 to 1.039] | 1.351 [1.060 to 1.722]
  Urine B2M, Week 48, n=119, 103: number analyzed (Participants) | 119 | 103
  Urine B2M, Week 48, n=119, 103 | 0.900 [0.792 to 1.022] | 1.338 [1.148 to 1.560]
  Urine Albumin/Creatinine, Week 24, n=254, 252: number analyzed (Participants) | 254 | 252
  Urine Albumin/Creatinine, Week 24, n=254, 252 | 1.014 [0.927 to 1.109] | 1.050 [0.964 to 1.144]
  Urine Albumin/Creatinine , Week 48, n=237, 244: number analyzed (Participants) | 237 | 244
  Urine Albumin/Creatinine , Week 48, n=237, 244 | 0.934 [0.857 to 1.017] | 1.048 [0.968 to 1.134]
  Urine B2M/Urine Creatinine, Week 24, n=121, 95: number analyzed (Participants) | 121 | 95
  Urine B2M/Urine Creatinine, Week 24, n=121, 95 | 0.852 [0.737 to 0.985] | 1.331 [1.071 to 1.655]
  Urine B2M/Urine Creatinine, Week 48, n=114, 100: number analyzed (Participants) | 114 | 100
  Urine B2M/Urine Creatinine, Week 48, n=114, 100 | 0.888 [0.777 to 1.015] | 1.278 [1.119 to 1.458]
  Urine Phosphate, Week 24, n=330, 332: number analyzed (Participants) | 330 | 332
  Urine Phosphate, Week 24, n=330, 332 | 1.115 [1.025 to 1.212] | 1.012 [0.934 to 1.095]
  Urine Phosphate, Week 48, n=316, 330: number analyzed (Participants) | 316 | 330
  Urine Phosphate, Week 48, n=316, 330 | 1.061 [0.983 to 1.145] | 1.075 [0.996 to 1.159]
  Urine Protein/Creatinine, Week 24, n=269, 265: number analyzed (Participants) | 269 | 265
  Urine Protein/Creatinine, Week 24, n=269, 265 | 0.850 [0.806 to 0.895] | 1.016 [0.960 to 1.075]
  Urine Protein/Creatinine, Week 48, n=252, 269: number analyzed (Participants) | 252 | 269
  Urine Protein/Creatinine, Week 48, n=252, 269 | 0.879 [0.838 to 0.922] | 1.061 [1.009 to 1.115]
  Urine RBP 4, Week 24, n=332, 330: number analyzed (Participants) | 332 | 330
  Urine RBP 4, Week 24, n=332, 330 | 0.934 [0.842 to 1.036] | 1.073 [0.951 to 1.209]
  Urine RBP 4, Week 48, n=318, 328: number analyzed (Participants) | 318 | 328
  Urine RBP 4, Week 48, n=318, 328 | 1.115 [1.009 to 1.233] | 1.490 [1.332 to 1.667]
  Urine RBP 4/Urine Creatinine, Week 24, n=329, 330: number analyzed (Participants) | 329 | 330
  Urine RBP 4/Urine Creatinine, Week 24, n=329, 330 | 0.919 [0.846 to 0.998] | 1.110 [1.003 to 1.228]
  Urine RBP 4/Urine Creatinine, Week 48, n=304, 318: number analyzed (Participants) | 304 | 318
  Urine RBP 4/Urine Creatinine, Week 48, n=304, 318 | 1.147 [1.060 to 1.241] | 1.500 [1.367 to 1.646]
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.915, 95% CI 2-sided [0.887 to 0.943] — Week 24. Serum B2M
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.904, 95% CI 2-sided [0.880 to 0.929] — Week 48. Serum B2M
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.005, Mixed Model Repeated Measures; Ratio of geometric means = 0.656, 95% CI 2-sided [0.491 to 0.877] — Week 24. Urine B2M
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.672, 95% CI 2-sided [0.551 to 0.821] — Week 48. Urine B2M
Statistical Analysis 5: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.575, Mixed Model Repeated Measures; Ratio of geometric means = 0.965, 95% CI 2-sided [0.853 to 1.092] — Week 24. Urine Albumin/Creatinine
Statistical Analysis 6: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.051, Mixed Model Repeated Measures; Ratio of geometric means = 0.891, 95% CI 2-sided [0.793 to 1.001] — Week 48. Urine Albumin/Creatinine
Statistical Analysis 7: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.640, 95% CI 2-sided [0.493 to 0.831] — Week 24. Urine B2M/Urine Creatinine
Statistical Analysis 8: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.695, 95% CI 2-sided [0.576 to 0.839] — Week 48. Urine B2M/Urine Creatinine
Statistical Analysis 9: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.099, Mixed Model Repeated Measures; Ratio of geometric means = 1.102, 95% CI 2-sided [0.982 to 1.237] — Week 24. Urine Phosphate
Statistical Analysis 10: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.816, Mixed Model Repeated Measures; Ratio of geometric means = 0.987, 95% CI 2-sided [0.886 to 1.100] — Week 48. Urine Phosphate
Statistical Analysis 11: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.836, 95% CI 2-sided [0.774 to 0.904] — Week 24. Urine Protein/Creatinine
Statistical Analysis 12: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.829, 95% CI 2-sided [0.773 to 0.888] — Week 48. Urine Protein/Creatinine
Statistical Analysis 13: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.087, Mixed Model Repeated Measures; Ratio of geometric means = 0.871, 95% CI 2-sided [0.743 to 1.020] — Week 24. Urine RBP 4
Statistical Analysis 14: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.748, 95% CI 2-sided [0.644 to 0.870] — Week 48. Urine RBP 4
Statistical Analysis 15: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.005, Mixed Model Repeated Measures; Ratio of geometric means = 0.828, 95% CI 2-sided [0.727 to 0.944] — Week 24. Urine RBP 4/Urine Creatinine
Statistical Analysis 16: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.765, 95% CI 2-sided [0.677 to 0.864] — Week 48. Urine RBP 4/Urine Creatinine

34. Secondary Outcome: Ratio to Baseline in Renal Biomarkers- Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine and Urine RBP 4/Urine Creatinine at Week 96
Description: Blood and/or urine were collected to perform evaluation of renal inflammation biomarkers which included Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine, Urine RBP 4 and Urine RBP 4/Urine Creatinine. Baseline value is defined as the latest pre-dose assessment (Day 1). Ratio to Baseline was calculated as ratio of post-dose visit value over Baseline value. Statistical analysis of changes from baseline were performed on log-transformed data. Results were transformed back via exponential transformation such that treatment comparisons are assessed via odds ratios. Estimated ratio of geometric means (each visit over Baseline) and 95% confidence interval (CI) have been presented.
Time Frame: Baseline (Day 1) and Week 96
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Ratio
  Urine Albumin/Creatinine, Week 96, n=222, 243: number analyzed (Participants) | 222 | 243
  Urine Albumin/Creatinine, Week 96, n=222, 243 | 0.924 [0.847 to 1.008] | 1.101 [1.008 to 1.202]
  Urine B2M/Urine Creatinine , Week 96, n=107, 104: number analyzed (Participants) | 107 | 104
  Urine B2M/Urine Creatinine , Week 96, n=107, 104 | 0.794 [0.720 to 0.877] | 1.441 [1.193 to 1.740]
  Urine Phosphate, Week 96, n=292, 316: number analyzed (Participants) | 292 | 316
  Urine Phosphate, Week 96, n=292, 316 | 1.113 [1.021 to 1.214] | 1.066 [0.984 to 1.155]
  Urine Protein/Creatinine, Week 96, n=238, 258: number analyzed (Participants) | 238 | 258
  Urine Protein/Creatinine, Week 96, n=238, 258 | 0.868 [0.818 to 0.920] | 1.053 [1.004 to 1.105]
  Urine RBP 4/Urine Creatinine, Week 96, n=289, 311: number analyzed (Participants) | 289 | 311
  Urine RBP 4/Urine Creatinine, Week 96, n=289, 311 | 1.310 [1.207 to 1.420] | 1.771 [1.604 to 1.955]
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.006, Mixed Model Repeated Measures; Ratio of geometric means = 0.839, 95% CI 2-sided [0.742 to 0.950] — Week 96. Urine Albumin/Creatinine
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.551, 95% CI 2-sided [0.445 to 0.682] — Week 96. Urine B2M/Urine Creatinine
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.467, Mixed Model Repeated Measures; Ratio of geometric means = 1.045, 95% CI 2-sided [0.928 to 1.175] — Week 96. Urine Phosphate
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.824, 95% CI 2-sided [0.764 to 0.889] — Week 96. Urine Protein/Creatinine
Statistical Analysis 5: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.740, 95% CI 2-sided [0.651 to 0.840] — Week 96. Urine RBP 4/Urine Creatinine

35. Secondary Outcome: Ratio to Baseline in Renal Biomarkers- Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine and Urine RBP 4/Urine Creatinine at Week 144
Description: as for outcome 33
Time Frame: Baseline (Day 1) and Week 144
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Ratio
  Urine Albumin/Creatinine , Week 144, n=207, 212: number analyzed (Participants) | 207 | 212
  Urine Albumin/Creatinine , Week 144, n=207, 212 | 1.050 [0.954 to 1.155] | 1.146 [1.039 to 1.264]
  Urine B2M/Urine Creatinine , Week 144, n=100, 102: number analyzed (Participants) | 100 | 102
  Urine B2M/Urine Creatinine , Week 144, n=100, 102 | 0.751 [0.679 to 0.830] | 1.518 [1.281 to 1.799]
  Urine Phosphate, Week 144, n=274, 294: number analyzed (Participants) | 274 | 294
  Urine Phosphate, Week 144, n=274, 294 | 1.040 [0.954 to 1.133] | 0.955 [0.879 to 1.037]
  Urine Protein/Creatinine , Week 144, n=225,232: number analyzed (Participants) | 225 | 232
  Urine Protein/Creatinine , Week 144, n=225,232 | 0.988 [0.932 to 1.047] | 1.210 [1.144 to 1.280]
  Urine RBP 4/Urine Creatinine, Week 144, n=276, 292: number analyzed (Participants) | 276 | 292
  Urine RBP 4/Urine Creatinine, Week 144, n=276, 292 | 1.648 [1.550 to 1.752] | 2.425 [2.208 to 2.663]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.205, Mixed Model Repeated Measures; Ratio of geometric means = 0.916, 95% CI 2-sided [0.799 to 1.050] — Week 144. Urine Albumin/Creatinine
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.495, 95% CI 2-sided [0.406 to 0.603] — Week 144. Urine B2M/Urine Creatinine
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.160, Mixed Model Repeated Measures; Ratio of geometric means = 1.089, 95% CI 2-sided [0.967 to 1.226] — Week 144. Urine Phosphate
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.817, 95% CI 2-sided [0.753 to 0.885] — Week 144. Urine Protein/Creatinine
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Ratio of geometric means = 0.679, 95% CI 2-sided [0.607 to 0.760] — Week 144. Urine RBP 4/Urine Creatinine

36. Secondary Outcome: Change From Baseline in Bone Biomarkers-Serum Bone Specific Alkaline Phosphatase (Bone-ALP), Serum Osteocalcin, Serum Procollagen 1 N-Terminal Propeptide (PINP) and Serum Type I Collagen C-Telopeptides (CTX-1) at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of bone biomarkers which included bone-ALP, Serum Osteocalcin, PINP and CTX-1. Baseline value is defined as the latest pre-dose assessment (Day 1). Change from Baseline was calculated as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, baseline plasma HIV-1 RNA (factor), baseline CD4+ cell count (factor), age, sex (factor), race (factor), BMI (factor), smoking status (factor), current Vitamin D use (factor), baseline biomarker value, treatment and visit interaction, and baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Micrograms per Liter (ug/L)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Micrograms per Liter (ug/L)
  Bone-ALP, Week 24, n=334, 332: number analyzed (Participants) | 334 | 332
  Bone-ALP, Week 24, n=334, 332 | 0.91 (0.179) | 3.13 (0.199)
  Bone-ALP, Week 48, n=321, 331: number analyzed (Participants) | 321 | 331
  Bone-ALP, Week 48, n=321, 331 | 1.21 (0.193) | 3.79 (0.239)
  Serum Osteocalcin, Week 24, n=335, 334: number analyzed (Participants) | 335 | 334
  Serum Osteocalcin, Week 24, n=335, 334 | 2.56 (0.341) | 6.74 (0.347)
  Serum Osteocalcin, Week 48, n=322, 330: number analyzed (Participants) | 322 | 330
  Serum Osteocalcin, Week 48, n=322, 330 | 0.78 (0.311) | 6.01 (0.400)
  PINP, Week 24, n=337, 336: number analyzed (Participants) | 337 | 336
  PINP, Week 24, n=337, 336 | 4.5 (0.91) | 18.3 (1.06)
  PINP, Week 48, n=321, 334: number analyzed (Participants) | 321 | 334
  PINP, Week 48, n=321, 334 | 0.5 (0.83) | 13.1 (0.84)
  CTX-1, Week 24, n=337, 334: number analyzed (Participants) | 337 | 334
  CTX-1, Week 24, n=337, 334 | 0.1192 (0.01304) | 0.2820 (0.01472)
  CTX-1, Week 48, n=323, 331: number analyzed (Participants) | 323 | 331
  CTX-1, Week 48, n=323, 331 | 0.1338 (0.01258) | 0.3352 (0.01885)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -2.23, 95% CI 2-sided [-2.75 to -1.70] — Week 24. Bone ALP
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -2.58, 95% CI 2-sided [-3.19 to -1.98] — Week 48. Bone ALP
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -4.19, 95% CI 2-sided [-5.15 to -3.23] — Week 28. Serum Osteocalcin
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -5.23, 95% CI 2-sided [-6.22 to -4.23] — Week 48. Serum Osteocalcin
Statistical Analysis 5: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -13.8, 95% CI 2-sided [-16.5 to -11.1] — Week 24. Serum PINP
Statistical Analysis 6: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -12.6, 95% CI 2-sided [-15.0 to -10.3] — Week 48. Serum PINP
Statistical Analysis 7: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -0.1628, 95% CI 2-sided [-0.2015 to -0.1241] — Week 24. CTX-1
Statistical Analysis 8: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -0.2015, 95% CI 2-sided [-0.2460 to -0.1569] — Week 48. CTX-1

37. Secondary Outcome: Change From Baseline in Bone Biomarkers-Serum Bone-ALP, Serum Osteocalcin, Serum PINP and Serum Type I CTX-1 at Week 96
Description: as for outcome 36
Time Frame: Baseline (Day 1) and at Week 96
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Micrograms per Liter (ug/L)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Micrograms per Liter (ug/L)
  Bone-ALP, Week 96, n=296, 317: number analyzed (Participants) | 296 | 317
  Bone-ALP, Week 96, n=296, 317 | 0.30 (0.191) | 2.37 (0.216)
  Serum Osteocalcin, Week 96, n=297, 320: number analyzed (Participants) | 297 | 320
  Serum Osteocalcin, Week 96, n=297, 320 | 0.40 (0.345) | 4.57 (0.391)
  PINP, Week 96, n=297, 319: number analyzed (Participants) | 297 | 319
  PINP, Week 96, n=297, 319 | 15.0 (1.63) | 28.3 (1.50)
  CTX-1, Week 96, n=297, 315: number analyzed (Participants) | 297 | 315
  CTX-1, Week 96, n=297, 315 | 0.1351 (0.01580) | 0.2943 (0.01916)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -2.06, 95% CI 2-sided [-2.63 to -1.50] — Week 96, Bone ALP
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -4.17, 95% CI 2-sided [-5.20 to -3.14] — Week 96, Serum Osteocalcin
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -13.3, 95% CI 2-sided [-17.6 to -8.9] — Week 96, Serum PINP
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -0.1592, 95% CI 2-sided [-0.2080 to -0.1104] — Week 96, CTX-1

38. Secondary Outcome: Change From Baseline in Bone Biomarkers-Serum Bone-ALP, Serum Osteocalcin, Serum PINP and Serum Type I CTX-1 at Week 144
Description: as for outcome 36
Time Frame: Baseline (Day 1) and at Week 144
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Micrograms per Liter (ug/L)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Micrograms per Liter (ug/L)
  Bone-ALP, Week 144, n=281, 295: number analyzed (Participants) | 281 | 295
  Bone-ALP, Week 144, n=281, 295 | -0.25 (0.172) | 1.43 (0.217)
  Serum Osteocalcin, Week 144, n=281, 299: number analyzed (Participants) | 281 | 299
  Serum Osteocalcin, Week 144, n=281, 299 | 0.29 (0.374) | 3.21 (0.403)
  PINP, Week 144, n=281,299: number analyzed (Participants) | 281 | 299
  PINP, Week 144, n=281,299 | 4.6 (1.04) | 13.8 (1.14)
  CTX-1, Week 144, n=281, 296: number analyzed (Participants) | 281 | 296
  CTX-1, Week 144, n=281, 296 | 0.0750 (0.01150) | 0.2164 (0.01407)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -1.68, 95% CI 2-sided [-2.23 to -1.14] — Week 144, Bone ALP
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -2.91, 95% CI 2-sided [-4.00 to -1.83] — Week 144, Serum Osteocalcin
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -9.2, 95% CI 2-sided [-12.3 to -6.2] — Week 144, Serum PINP
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -0.1414, 95% CI 2-sided [-0.1771 to -0.1056] — Week 144, CTX-1

39. Secondary Outcome: Change From Baseline in Bone Biomarker-Serum Vitamin D at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of bone biomarker serum vitamin D. Baseline value is defined as the latest pre-dose assessment (Day 1). Change from Baseline was calculated as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, baseline plasma HIV-1 RNA (factor), baseline CD4+ cell count (factor), age, sex (factor), race (factor), BMI (factor), smoking status (factor), current Vitamin D use (factor), baseline biomarker value, treatment and visit interaction, and baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Nanomoles per Liter (nmol/L)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Nanomoles per Liter (nmol/L)
  Serum Vitamin D, Week 24, n=337, 337: number analyzed (Participants) | 337 | 337
  Serum Vitamin D, Week 24, n=337, 337 | 5.9 (1.15) | 12.4 (1.33)
  Serum Vitamin D, Week 48, n=322, 333: number analyzed (Participants) | 322 | 333
  Serum Vitamin D, Week 48, n=322, 333 | -3.1 (0.89) | 3.1 (1.10)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -6.5, 95% CI 2-sided [-9.9 to -3.0] — Week 24
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p < 0.001, Mixed Model Repeated Measures; Mean Difference (Net) = -6.2, 95% CI 2-sided [-9.0 to -3.4] — Week 48

40. Secondary Outcome: Change From Baseline in Bone Biomarker-Serum Vitamin D at Week 96
Description: as for outcome 39
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Nanomoles per Liter (nmol/L)
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 298 | 320
Nanomoles per Liter (nmol/L) | -2.2 (1.05) | 0.7 (1.04)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.048, Mixed Model Repeated Measures; Mean Difference (Net) = -2.9, 95% CI 2-sided [-5.8 to 0.0] — Week 96

41. Secondary Outcome: Change From Baseline in Bone Biomarker-Serum Vitamin D at Week 144
Description: as for outcome 39
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Nanomoles per Liter (nmol/L)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 281 | 298
Nanomoles per Liter (nmol/L) | -2.0 (1.16) | 2.9 (1.28)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.004, Mixed Model Repeated Measures; Mean Difference (Net) = -4.9, 95% CI 2-sided [-8.3 to -1.6] — Week 144

42. Secondary Outcome: Percentage Change From Baseline in Fasting Lipids-Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of fasting lipids which included Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides. Baseline value is defined as the latest pre-dose assessment (Day 1). Percentage change from Baseline was calculated as 100 multiplied by ([post-dose visit value minus Baseline value] divided by Baseline value).
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage change
  Serum or Plasma Cholesterol, Week 24, n=294, 297: number analyzed (Participants) | 294 | 297
  Serum or Plasma Cholesterol, Week 24, n=294, 297 | 9.4 (17.44) | -4.7 (16.12)
  Serum or Plasma Cholesterol, Week 48, n=280, 289: number analyzed (Participants) | 280 | 289
  Serum or Plasma Cholesterol, Week 48, n=280, 289 | 10.5 (18.89) | -2.4 (17.14)
  HDL Cholesterol, Direct, Week 24, n=294, 297: number analyzed (Participants) | 294 | 297
  HDL Cholesterol, Direct, Week 24, n=294, 297 | 16.4 (22.58) | 3.4 (21.55)
  HDL Cholesterol, Direct, Week 48, n=280, 289: number analyzed (Participants) | 280 | 289
  HDL Cholesterol, Direct, Week 48, n=280, 289 | 15.0 (25.07) | 5.0 (33.04)
  LDL Cholesterol, Week 24, n=294, 297: number analyzed (Participants) | 294 | 297
  LDL Cholesterol, Week 24, n=294, 297 | 12.4 (45.05) | -8.1 (23.70)
  LDL Cholesterol, Week 48, n=280, 289: number analyzed (Participants) | 280 | 289
  LDL Cholesterol, Week 48, n=280, 289 | 14.8 (48.74) | -4.0 (24.06)
  Triglycerides ,Week 24, n=294, 297: number analyzed (Participants) | 294 | 297
  Triglycerides ,Week 24, n=294, 297 | 8.5 (46.57) | 4.3 (72.35)
  Triglycerides , Week 48, n=280, 289: number analyzed (Participants) | 280 | 289
  Triglycerides , Week 48, n=280, 289 | 12.8 (68.99) | 4.4 (70.43)

43. Secondary Outcome: Change From Baseline in Fasting Lipids-Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides at Week 96
Description: Blood samples were collected to perform evaluation of fasting lipids which included Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides. Baseline value was defined as the latest pre-dose assessment (Day 1). Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Error); unit: Millimoles per liter
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 253 | 277
Millimoles per liter
  Serum or Plasma Cholesterol, Week 96 | 0.379 (0.0376) | -0.104 (0.0378)
  HDL Cholesterol, Direct, Week 96 | 0.199 (0.0156) | 0.090 (0.0149)
  LDL Cholesterol, Week 96, | 0.147 (0.0338) | -0.154 (0.0303)
  Triglycerides, Week 96, | 0.129 (0.0835) | -0.112 (0.0358)

44. Secondary Outcome: Change From Baseline in Fasting Lipids-Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides at Week 144
Description: as for outcome 43
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Error); unit: Millimoles per liter
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 245 | 256
Millimoles per liter
  Serum or Plasma Cholesterol, Week 144, | 0.367 (0.0408) | -0.037 (0.0406)
  HDL Cholesterol, Direct, Week 144 | 0.181 (0.0150) | 0.098 (0.0147)
  LDL Cholesterol, Week 144, | 0.170 (0.0336) | -0.105 (0.0348)
  Triglycerides, Week 144 | 0.117 (0.0872) | -0.104 (0.0385)

45. Secondary Outcome: Percentage Change From Baseline in Fasting Lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of fasting lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio. Baseline value is the latest pre-dose assessment (Day 1). Percentage change from Baseline was calculated as 100 multiplied by ([post-dose visit value minus Baseline value] divided by Baseline value).
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage change
  Total/HDL Cholesterol Ratio, Week 24, n=294, 297: number analyzed (Participants) | 294 | 297
  Total/HDL Cholesterol Ratio, Week 24, n=294, 297 | -4.0 (19.08) | -4.6 (27.52)
  Total/HDL Cholesterol Ratio, Week 48, n=280, 289: number analyzed (Participants) | 280 | 289
  Total/HDL Cholesterol Ratio, Week 48, n=280, 289 | -0.2 (31.10) | -4.4 (16.96)

46. Secondary Outcome: Change From Baseline in Fasting Lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio at Week 96
Description: Blood samples were collected to perform evaluation of fasting lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio. Baseline value was defined as the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error has been presented.
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 253 | 277
Ratio | -0.213 (0.0566) | -0.402 (0.0479)

47. Secondary Outcome: Change From Baseline in Fasting Lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio at Week 144
Description: as for outcome 46
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 245 | 256
Ratio | -0.229 (0.0559) | -0.386 (0.0463)

48. Secondary Outcome: Percentage of Participants With Grade 2 or Greater Laboratory Abnormalities in Fasting LDL Cholesterol by Weeks 24, 48
Description: Blood samples were collected to perform evaluation of fasting LDL cholesterol. Any abnormalities were evaluated by the investigator and graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Percentage of participants with Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Weeks 24 and 48 have been presented. Participants without any post-Baseline fasting LDL cholesterol value prior to Week 48 or those who had Baseline lipids-lowering agents are not included. Lipid Last Observation Carried Forward (LOCF) data was used such that the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering agent was used in place of future observed values. Percentage values are rounded to the nearest whole digit.
Time Frame: Weeks 24 and Week 48
Population: as for outcome 22
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants
  Week 24, n=309, 316: number analyzed (Participants) | 309 | 316
  Week 24, n=309, 316 | 4 | 2
  Week 48, n=318, 320: number analyzed (Participants) | 318 | 320
  Week 48, n=318, 320 | 4 | 3
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.157, Fisher Exact — Fisher's exact p-value; Difference in percentage = 2.0, 95% CI 2-sided [-0.6 to 4.6] — Week 24
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.414, Fisher Exact — Fisher's exact p-value; Difference in percentage = 1.3, 95% CI 2-sided [-1.7 to 4.2] — Week 48

49. Secondary Outcome: Percentage of Participants With Grade 2 or Greater Laboratory Abnormalities in Fasting LDL Cholesterol by Week 96
Description: Blood samples were collected to perform evaluation of fasting LDL cholesterol. Any abnormalities were evaluated by the investigator and graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Percentage of participants with Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Week 96 have been presented. Participants without any post-Baseline fasting LDL cholesterol value prior to Week 96 or those who had Baseline lipids-lowering agents were not included. Lipid Last Observation Carried Forward (LOCF) data was used such that the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering agent was used in place of future observed values. Percentage values are rounded to the nearest whole digit.
Time Frame: Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 320 | 323
Percentage of participants | 5 | 4
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.562, Fisher Exact — Fisher's exact p-value; Difference in percentage = 1.0, 95% CI 2-sided [-2.1 to 4.1] — Week 96

50. Secondary Outcome: Percentage of Participants With Grade 2 or Greater Laboratory Abnormalities in Fasting LDL Cholesterol by Week 144
Description: Blood samples were collected to perform evaluation of fasting LDL cholesterol. Any abnormalities were evaluated by the investigator and graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). Percentage of participants with Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Week 144 have been presented. Participants without any post-Baseline fasting LDL cholesterol value prior to Week 144 or those who had Baseline lipids-lowering agents were not included. Lipid Last Observation Carried Forward (LOCF) data was used such that the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering agent was used in place of future observed values. Percentage values are rounded to the nearest whole digit.
Time Frame: Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 321 | 322
Percentage of participants | 5 | 4
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.587, Fisher Exact — Fisher's exact p-value; Difference in percentage = 0.9, 95% CI 2-sided [-2.4 to 4.3] — Week 144

51. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count, Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 24
Description: Percentage of participants by subgroups (by age, gender, Baseline CD4+ cell count, Baseline HIV-1 RNA, race) with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. Data was presented by subgroups: age (<35, 35 to <50, >=50 years); gender (males and females), Baseline CD4+ cell count (<=200, >200), Baseline HIV-1 RNA (<=100000, >100000) and Race (White, African American/African H., Asian, Other). Percentage values are rounded to the nearest whole digit.
Time Frame: Week 24
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants
  Baseline CD4+ cell count, <=200,n=31,29: number analyzed (Participants) | 31 | 29
  Baseline CD4+ cell count, <=200,n=31,29 | 90 | 86
  Baseline CD4+ cell count, >200,n=325,329: number analyzed (Participants) | 325 | 329
  Baseline CD4+ cell count, >200,n=325,329 | 93 | 94
  Female, n=59, 52: number analyzed (Participants) | 59 | 52
  Female, n=59, 52 | 93 | 96
  Male, n=297, 306: number analyzed (Participants) | 297 | 306
  Male, n=297, 306 | 92 | 92
  Age, <35,n= 211, 205: number analyzed (Participants) | 211 | 205
  Age, <35,n= 211, 205 | 93 | 95
  Age, 35 to <50,n=116, 107: number analyzed (Participants) | 116 | 107
  Age, 35 to <50,n=116, 107 | 91 | 93
  Age, >=50, n=29, 46: number analyzed (Participants) | 29 | 46
  Age, >=50, n=29, 46 | 93 | 85
  Baseline plasma HIV-1 RNA, <=100000,n=282,282: number analyzed (Participants) | 282 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=282,282 | 93 | 95
  Baseline plasma HIV-1 RNA, >100000,n=74, 76: number analyzed (Participants) | 74 | 76
  Baseline plasma HIV-1 RNA, >100000,n=74, 76 | 92 | 87
  Race, White, n=244,247: number analyzed (Participants) | 244 | 247
  Race, White, n=244,247 | 93 | 95
  Race, African American/African H., n=39, 36: number analyzed (Participants) | 39 | 36
  Race, African American/African H., n=39, 36 | 92 | 81
  Race, Asian, n=37, 42: number analyzed (Participants) | 37 | 42
  Race, Asian, n=37, 42 | 89 | 93
  Race, Other, n=36, 33: number analyzed (Participants) | 36 | 33
  Race, Other, n=36, 33 | 94 | 94

52. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 48
Description: as for outcome 51
Time Frame: Week 48
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants
  Baseline CD4+ cell count, <=200,n=31,29: number analyzed (Participants) | 31 | 29
  Baseline CD4+ cell count, <=200,n=31,29 | 81 | 90
  Baseline CD4+ cell count, >200,n=325,329: number analyzed (Participants) | 325 | 329
  Baseline CD4+ cell count, >200,n=325,329 | 91 | 93
  Female, n=59, 52: number analyzed (Participants) | 59 | 52
  Female, n=59, 52 | 88 | 94
  Male, n=297, 306: number analyzed (Participants) | 297 | 306
  Male, n=297, 306 | 90 | 92
  Age, <35,n= 211, 205: number analyzed (Participants) | 211 | 205
  Age, <35,n= 211, 205 | 92 | 93
  Age, 35 to <50,n=116, 107: number analyzed (Participants) | 116 | 107
  Age, 35 to <50,n=116, 107 | 86 | 94
  Age, >=50, n=29, 46: number analyzed (Participants) | 29 | 46
  Age, >=50, n=29, 46 | 90 | 87
  Baseline plasma HIV-1 RNA, <=100000,n=282,282: number analyzed (Participants) | 282 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=282,282 | 90 | 93
  Baseline plasma HIV-1 RNA, >100000,n=74, 76: number analyzed (Participants) | 74 | 76
  Baseline plasma HIV-1 RNA, >100000,n=74, 76 | 88 | 91
  Race, White, n=244,247: number analyzed (Participants) | 244 | 247
  Race, White, n=244,247 | 90 | 94
  Race, African American/African H., n=39, 36: number analyzed (Participants) | 39 | 36
  Race, African American/African H., n=39, 36 | 87 | 81
  Race, Asian, n=37, 42: number analyzed (Participants) | 37 | 42
  Race, Asian, n=37, 42 | 92 | 98
  Race, Other, n=36, 33: number analyzed (Participants) | 36 | 33
  Race, Other, n=36, 33 | 89 | 94

53. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 96
Description: Percentage of participants by subgroups (by age, gender, Baseline CD4+ cell count, Baseline HIV-1 RNA, race) with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. Data was presented by subgroups: age (<35, 35 to <50, >=50 years); gender (males and females), Baseline CD4+ cell count (<=200 cells/mm^3, >200 cells/mm^3), Baseline HIV-1 RNA (<=100000, >100000) and Race (White, African American/African H., Asian and other). Percentage values are rounded to the nearest whole digit.
Time Frame: Week 96
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants
  Baseline CD4+ cell count, <=200,n=31, 29: number analyzed (Participants) | 31 | 29
  Baseline CD4+ cell count, <=200,n=31, 29 | 65 | 90
  Baseline CD4+ cell count, >200,n=325,329: number analyzed (Participants) | 325 | 329
  Baseline CD4+ cell count, >200,n=325,329 | 86 | 89
  Female, n=59, 52: number analyzed (Participants) | 59 | 52
  Female, n=59, 52 | 83 | 88
  Male, n=297,306,: number analyzed (Participants) | 297 | 306
  Male, n=297,306, | 85 | 90
  Age, <35,n= 211, 205: number analyzed (Participants) | 211 | 205
  Age, <35,n= 211, 205 | 84 | 90
  Age, 35 to <50,n=116, 107: number analyzed (Participants) | 116 | 107
  Age, 35 to <50,n=116, 107 | 84 | 89
  Age, >=50, n=29,46: number analyzed (Participants) | 29 | 46
  Age, >=50, n=29,46 | 86 | 87
  Baseline plasma HIV-1 RNA, <=100000,n=282,282: number analyzed (Participants) | 282 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=282,282 | 85 | 90
  Baseline plasma HIV-1 RNA, >100000,n=74, 76: number analyzed (Participants) | 74 | 76
  Baseline plasma HIV-1 RNA, >100000,n=74, 76 | 81 | 88
  Race, White, n=244,247: number analyzed (Participants) | 244 | 247
  Race, White, n=244,247 | 86 | 90
  Race, African American/African H., n=39,36: number analyzed (Participants) | 39 | 36
  Race, African American/African H., n=39,36 | 79 | 81
  Race, Asian, n=37, 42: number analyzed (Participants) | 37 | 42
  Race, Asian, n=37, 42 | 78 | 90
  Race, Other, n=36, 33: number analyzed (Participants) | 36 | 33
  Race, Other, n=36, 33 | 86 | 91

54. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 144
Description: as for outcome 53
Time Frame: Week 144
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Percentage of participants
  Baseline CD4+ cell count, <=200,n=31, 29: number analyzed (Participants) | 31 | 29
  Baseline CD4+ cell count, <=200,n=31, 29 | 58 | 83
  Baseline CD4+ cell count, >200,n=325,329: number analyzed (Participants) | 325 | 329
  Baseline CD4+ cell count, >200,n=325,329 | 81 | 83
  Female, n=59, 52: number analyzed (Participants) | 59 | 52
  Female, n=59, 52 | 71 | 85
  Male, n=297,306,: number analyzed (Participants) | 297 | 306
  Male, n=297,306, | 80 | 82
  Age, <35,n= 211, 205: number analyzed (Participants) | 211 | 205
  Age, <35,n= 211, 205 | 77 | 83
  Age, 35 to <50,n=116, 107: number analyzed (Participants) | 116 | 107
  Age, 35 to <50,n=116, 107 | 81 | 83
  Age, >=50, n=29,46: number analyzed (Participants) | 29 | 46
  Age, >=50, n=29,46 | 83 | 78
  Baseline plasma HIV-1 RNA, <=100000,n=282,282: number analyzed (Participants) | 282 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=282,282 | 79 | 82
  Baseline plasma HIV-1 RNA, >100000,n=74, 76: number analyzed (Participants) | 74 | 76
  Baseline plasma HIV-1 RNA, >100000,n=74, 76 | 78 | 87
  Race, White, n=244,247: number analyzed (Participants) | 244 | 247
  Race, White, n=244,247 | 82 | 85
  Race, African American/African H., n=39,36: number analyzed (Participants) | 39 | 36
  Race, African American/African H., n=39,36 | 69 | 72
  Race, Asian, n=37, 42: number analyzed (Participants) | 37 | 42
  Race, Asian, n=37, 42 | 73 | 81
  Race, Other, n=36, 33: number analyzed (Participants) | 36 | 33
  Race, Other, n=36, 33 | 78 | 79

55. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 24 by Subgroups
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented for subgroups (Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, Age, Gender, and race). For each subgroup, adjusted mean is the estimated mean change from Baseline in each arm calculated from ANCOVA model adjusting for the following covariates/factors: treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, subgroup, and treatment and relevant subgroup interaction. For CD4+ cell count subgroup, Baseline CD4+ cell count group is included as a factor only.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells per cubic millimeter
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Cells per cubic millimeter
  Baseline plasma HIV-1 RNA,<=100000, n=268,268: number analyzed (Participants) | 268 | 268
  Baseline plasma HIV-1 RNA,<=100000, n=268,268 | 187.72 (10.860) | 167.93 (10.842)
  Baseline plasma HIV-1 RNA,>100000, n=72,73: number analyzed (Participants) | 72 | 73
  Baseline plasma HIV-1 RNA,>100000, n=72,73 | 206.63 (21.107) | 205.96 (20.990)
  Baseline CD4+ cell count,<=200, n=29,27: number analyzed (Participants) | 29 | 27
  Baseline CD4+ cell count,<=200, n=29,27 | 157.01 (33.113) | 120.17 (34.151)
  Baseline CD4+ cell count,>200, n=311, 314: number analyzed (Participants) | 311 | 314
  Baseline CD4+ cell count,>200, n=311, 314 | 195.11 (10.026) | 180.73 (9.972)
  Age, <35,n= 203,199: number analyzed (Participants) | 203 | 199
  Age, <35,n= 203,199 | 202.76 (12.456) | 177.62 (12.563)
  Age, 35 to <50, n=109, 100: number analyzed (Participants) | 109 | 100
  Age, 35 to <50, n=109, 100 | 172.05 (16.983) | 179.87 (17.733)
  Age, >=50, n=28, 42: number analyzed (Participants) | 28 | 42
  Age, >=50, n=28, 42 | 188.79 (33.534) | 159.34 (27.344)
  Female, n=57,50: number analyzed (Participants) | 57 | 50
  Female, n=57,50 | 199.45 (23.498) | 181.78 (25.263)
  Male, n=283,291: number analyzed (Participants) | 283 | 291
  Male, n=283,291 | 190.21 (10.538) | 175.05 (10.400)
  Race, White, n=236,235: number analyzed (Participants) | 236 | 235
  Race, White, n=236,235 | 204.78 (11.531) | 182.27 (11.582)
  Race, African Am/African H., n=36,33: number analyzed (Participants) | 36 | 33
  Race, African Am/African H., n=36,33 | 143.84 (29.541) | 170.51 (30.870)
  Race, Asian, n=34, 41: number analyzed (Participants) | 34 | 41
  Race, Asian, n=34, 41 | 169.80 (30.491) | 165.36 (27.782)
  Race, Other, n=34,32: number analyzed (Participants) | 34 | 32
  Race, Other, n=34,32 | 174.30 (30.375) | 149.34 (31.404)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 19.80, 95% CI 2-sided [-10.23 to 49.83] — Baseline plasma HIV-1 RNA,<=100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, and treatment and HIV-1 RNA interaction
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 0.67, 95% CI 2-sided [-57.07 to 58.40] — Baseline plasma HIV-1 RNA,>100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, and treatment and HIV-1 RNA interaction
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 36.84, 95% CI 2-sided [-55.94 to 129.63] — Baseline CD4+ cell count,<=200. Following covariates were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, and treatment and Baseline CD4+ cell count interaction
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 14.37, 95% CI 2-sided [-13.38 to 42.12] — Baseline CD4+ cell count,>200. Following covariates were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, and treatment and Baseline CD4+ cell count interaction
Statistical Analysis 5: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 25.14, 95% CI 2-sided [-9.56 to 59.85] — Age<35. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 6: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -7.82, 95% CI 2-sided [-55.98 to 40.34] — Age 35 to <50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 7: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 29.45, 95% CI 2-sided [-55.47 to 114.38] — Age>=50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 8: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 17.67, 95% CI 2-sided [-49.89 to 85.23] — Female. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, gender, and treatment and gender interaction
Statistical Analysis 9: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 15.16, 95% CI 2-sided [-13.90 to 44.21] — Male. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, gender, and treatment and gender interaction
Statistical Analysis 10: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 22.51, 95% CI 2-sided [-9.52 to 54.54] — Race group white. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race group, and treatment and race group interaction
Statistical Analysis 11: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -26.67, 95% CI 2-sided [-110.64 to 57.30] — Race group African Am/African H.. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race group, and treatment and race group interaction
Statistical Analysis 12: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 4.44, 95% CI [-76.18 to 85.06] — Race group Asian. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race group, and treatment and race group interaction
Statistical Analysis 13: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 24.96, 95% CI 2-sided [-60.68 to 110.59] — Race group Other. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race group, and treatment and race group interaction

56. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 48 by Subgroups
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as post-dose visit value minus Baseline value. Adjusted mean and standard error is presented for subgroups (Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, Age group, Gender and race). For each subgroup, adjusted mean is the estimated mean change from Baseline in each arm calculated from Analysis of Covariance (ANCOVA) model adjusting for the following covariates/factors: treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, subgroup, and treatment and relevant subgroup interaction. For CD4+ cell count subgroup, Baseline CD4+ cell count group is included as a factor only.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells per cubic millimeter
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Cells per cubic millimeter
  Baseline plasma HIV-1 RNA,<=100000, n=257,264: number analyzed (Participants) | 257 | 264
  Baseline plasma HIV-1 RNA,<=100000, n=257,264 | 220.0 (11.72) | 212.4 (11.56)
  Baseline plasma HIV-1 RNA,>100000, n=67,70: number analyzed (Participants) | 67 | 70
  Baseline plasma HIV-1 RNA,>100000, n=67,70 | 238.5 (23.09) | 235.5 (22.70)
  Baseline CD4+ cell count,<=200, n=26, 27: number analyzed (Participants) | 26 | 27
  Baseline CD4+ cell count,<=200, n=26, 27 | 200.5 (36.97) | 177.9 (36.18)
  Baseline CD4+ cell count,>200, n=298, 307: number analyzed (Participants) | 298 | 307
  Baseline CD4+ cell count,>200, n=298, 307 | 225.9 (10.84) | 220.7 (10.68)
  Age group-1, <35,n= 194, 192: number analyzed (Participants) | 194 | 192
  Age group-1, <35,n= 194, 192 | 233.6 (13.49) | 225.2 (13.53)
  Age group-1, 35 to <50, n=104, 101: number analyzed (Participants) | 104 | 101
  Age group-1, 35 to <50, n=104, 101 | 208.7 (18.40) | 211.2 (18.67)
  Age group-1, >=50, n=26, 41: number analyzed (Participants) | 26 | 41
  Age group-1, >=50, n=26, 41 | 212.6 (36.84) | 194.8 (29.27)
  Female, n=54, 49: number analyzed (Participants) | 54 | 49
  Female, n=54, 49 | 237.1 (25.53) | 226.8 (26.98)
  Male, n=270, 285: number analyzed (Participants) | 270 | 285
  Male, n=270, 285 | 221.2 (11.41) | 215.6 (11.11)
  Race, White, n=224, 231: number analyzed (Participants) | 224 | 231
  Race, White, n=224, 231 | 226.0 (12.55) | 219.7 (12.39)
  Race, African Am/African H., n=33, 31: number analyzed (Participants) | 33 | 31
  Race, African Am/African H., n=33, 31 | 209.4 (32.75) | 239.9 (33.79)
  Race, Asian, n=34, 41: number analyzed (Participants) | 34 | 41
  Race, Asian, n=34, 41 | 246.4 (32.35) | 197.2 (29.47)
  Race, Other, n=33, 31: number analyzed (Participants) | 33 | 31
  Race, Other, n=33, 31 | 200.2 (32.69) | 202.7 (33.83)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 7.6, 95% CI 2-sided [-24.6 to 39.8] — Baseline plasma HIV-1 RNA,<=100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count and treatment and HIV-1 RNA interaction
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 3.0, 95% CI 2-sided [-59.8 to 65.9] — Baseline plasma HIV-1 RNA,>100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count and treatment and HIV-1 RNA interaction
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 22.6, 95% CI 2-sided [-78.3 to 123.5] — [estimate comment as in outcome 55, analysis 3]
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 5.2, 95% CI 2-sided [-24.7 to 35.1] — [estimate comment as in outcome 55, analysis 4]
Statistical Analysis 5: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 8.4, 95% CI 2-sided [-29.1 to 45.9] — [estimate comment as in outcome 55, analysis 5]
Statistical Analysis 6: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -2.5, 95% CI 2-sided [-53.9 to 48.9] — [estimate comment as in outcome 55, analysis 6]
Statistical Analysis 7: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 17.7, 95% CI 2-sided [-74.6 to 110.1] — [estimate comment as in outcome 55, analysis 7]
Statistical Analysis 8: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 10.4, 95% CI 2-sided [-62.3 to 83.1] — [estimate comment as in outcome 55, analysis 8]
Statistical Analysis 9: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 5.6, 95% CI 2-sided [-25.6 to 36.9] — [estimate comment as in outcome 55, analysis 9]
Statistical Analysis 10: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 6.3, 95% CI 2-sided [-28.2 to 40.9] — [estimate comment as in outcome 55, analysis 10]
Statistical Analysis 11: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -30.2, 95% CI 2-sided [-122.7 to 62.4] — [estimate comment as in outcome 55, analysis 11]
Statistical Analysis 12: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 49.2, 95% CI 2-sided [-36.3 to 134.7] — [estimate comment as in outcome 55, analysis 12]
Statistical Analysis 13: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -2.5, 95% CI 2-sided [-94.7 to 89.7] — [estimate comment as in outcome 55, analysis 13]

57. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 96 by Subgroups
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is the the latest pre-dose assessment (Day 1). Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted mean and standard error is presented for subgroups (Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, Age group, Gender and race). For each subgroup, adjusted mean is the estimated mean change from Baseline in each arm calculated from ANCOVA model adjusting for the following covariates/factors: treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, subgroup, and treatment and relevant subgroup interaction. For CD4+ cell count subgroup, Baseline CD4+ cell count group is included as a factor only.
Time Frame: Baseline (Day 1) and Week 96
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells per cubic millimeter
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Cells per cubic millimeter
  Baseline plasma HIV-1 RNA,<=100000, n=240,253: number analyzed (Participants) | 240 | 253
  Baseline plasma HIV-1 RNA,<=100000, n=240,253 | 254.8 (13.30) | 252.9 (12.93)
  Baseline plasma HIV-1 RNA,>100000, n=61,67: number analyzed (Participants) | 61 | 67
  Baseline plasma HIV-1 RNA,>100000, n=61,67 | 300.2 (26.50) | 260.1 (25.42)
  Baseline CD4+ cell count,<=200, n=21,26: number analyzed (Participants) | 21 | 26
  Baseline CD4+ cell count,<=200, n=21,26 | 240.5 (45.16) | 244.4 (40.44)
  Baseline CD4+ cell count,>200, n=280,294: number analyzed (Participants) | 280 | 294
  Baseline CD4+ cell count,>200, n=280,294 | 265.9 (12.28) | 255.1 (11.98)
  Age group-1, <35,n= 179,185: number analyzed (Participants) | 179 | 185
  Age group-1, <35,n= 179,185 | 270.2 (15.38) | 263.0 (15.09)
  Age group-1, 35 to <50, n=97,95: number analyzed (Participants) | 97 | 95
  Age group-1, 35 to <50, n=97,95 | 259.5 (20.86) | 262.0 (21.09)
  Age group-1, >=50, n=25, 40: number analyzed (Participants) | 25 | 40
  Age group-1, >=50, n=25, 40 | 237.6 (41.11) | 195.9 (32.45)
  Female, n=49,46: number analyzed (Participants) | 49 | 46
  Female, n=49,46 | 277.9 (29.40) | 259.1 (30.54)
  Male, n=252, 274: number analyzed (Participants) | 252 | 274
  Male, n=252, 274 | 261.4 (12.95) | 253.5 (12.43)
  Race group, White, n=210,223: number analyzed (Participants) | 210 | 223
  Race group, White, n=210,223 | 275.2 (14.21) | 260.0 (13.80)
  Race group, African Am/African H., n=31,29: number analyzed (Participants) | 31 | 29
  Race group, African Am/African H., n=31,29 | 228.5 (37.07) | 230.2 (38.23)
  Race group, Asian, n=29,38: number analyzed (Participants) | 29 | 38
  Race group, Asian, n=29,38 | 212.1 (38.34) | 244.8 (33.53)
  Race group, Other, n=31,30: number analyzed (Participants) | 31 | 30
  Race group, Other, n=31,30 | 273.4 (36.97) | 247.3 (37.67)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 1.9, 95% CI 2-sided [-34.5 to 38.2] — Baseline plasma HIV-1 RNA,<=100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, Baseline plasma HIV-1 RNA, and treatment and relevant Baseline plasma HIV-1 RNA interaction
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 40.1, 95% CI 2-sided [-31.2 to 111.5] — [estimate comment as in outcome 55, analysis 2]
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -3.9, 95% CI 2-sided [-122.3 to 114.5] — [estimate comment as in outcome 55, analysis 3]
Statistical Analysis 4: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 10.8, 95% CI 2-sided [-22.9 to 44.5] — [estimate comment as in outcome 55, analysis 4]
Statistical Analysis 5: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 7.3, 95% CI 2-sided [-35.0 to 49.6] — Age Group,<35. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 6: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -2.5, 95% CI 2-sided [-60.7 to 55.7] — Age Group,35 to <50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 7: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 41.6, 95% CI 2-sided [-61.2 to 144.5] — [estimate comment as in outcome 55, analysis 7]
Statistical Analysis 8: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 18.8, 95% CI 2-sided [-64.2 to 101.8] — [estimate comment as in outcome 55, analysis 8]
Statistical Analysis 9: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 7.8, 95% CI 2-sided [-27.4 to 43.1] — [estimate comment as in outcome 55, analysis 9]
Statistical Analysis 10: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 15.2, 95% CI 2-sided [-23.6 to 54.0] — Race group-white. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction
Statistical Analysis 11: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = -1.7, 95% CI 2-sided [-106.3 to 103.0] — Race group-African Am/African H. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction
Statistical Analysis 12: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Median Difference (Net) = -32.6, 95% CI 2-sided [-132.2 to 66.9] — Race group-Asian. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction
Statistical Analysis 13: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; Mean Difference (Net) = 26.1, 95% CI 2-sided [-77.3 to 129.5] — Race group-Other. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction

58. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 144 by Subgroups
Description: as for outcome 57
Time Frame: Baseline (Day 1) and Week 144
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells per cubic millimeter
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 356 | 358
Cells per cubic millimeter
  Baseline plasma HIV-1 RNA,<=100000, n=214,223: number analyzed (Participants) | 214 | 223
  Baseline plasma HIV-1 RNA,<=100000, n=214,223 | 295.7 (14.14) | 296.1 (13.84)
  Baseline plasma HIV-1 RNA,>100000, n=56, 64: number analyzed (Participants) | 56 | 64
  Baseline plasma HIV-1 RNA,>100000, n=56, 64 | 334.3 (27.77) | 329.6 (26.15)
  Baseline CD4+ cell count,<=200, n=17, 24: number analyzed (Participants) | 17 | 24
  Baseline CD4+ cell count,<=200, n=17, 24 | 290.2 (50.44) | 272.9 (42.29)
  Baseline CD4+ cell count,>200, n=253, 263: number analyzed (Participants) | 253 | 263
  Baseline CD4+ cell count,>200, n=253, 263 | 304.7 (12.97) | 306.2 (12.71)
  Age group, <35,n=155, 167: number analyzed (Participants) | 155 | 167
  Age group, <35,n=155, 167 | 298.0 (16.59) | 316.0 (15.93)
  Age group-1, 35 to <50, n=92, 87: number analyzed (Participants) | 92 | 87
  Age group-1, 35 to <50, n=92, 87 | 305.6 (21.48) | 302.1 (22.11)
  Age group-1, >=50, n=23,33: number analyzed (Participants) | 23 | 33
  Age group-1, >=50, n=23,33 | 337.4 (43.01) | 242.2 (35.83)
  Female, n=43, 43: number analyzed (Participants) | 43 | 43
  Female, n=43, 43 | 346.6 (31.40) | 321.7 (31.67)
  Male, n=227, 244: number analyzed (Participants) | 227 | 244
  Male, n=227, 244 | 295.9 (13.66) | 300.0 (13.20)
  Race group, White, n=190,201: number analyzed (Participants) | 190 | 201
  Race group, White, n=190,201 | 314.2 (14.93) | 314.0 (14.53)
  Race group, African Am/African H., n=26, 26: number analyzed (Participants) | 26 | 26
  Race group, African Am/African H., n=26, 26 | 243.8 (40.42) | 295.1 (40.39)
  Race group, Asian, n=26, 34: number analyzed (Participants) | 26 | 34
  Race group, Asian, n=26, 34 | 244.0 (40.47) | 264.1 (35.41)
  Race group, Other, n=28,26: number analyzed (Participants) | 28 | 26
  Race group, Other, n=28,26 | 346.2 (38.87) | 279.9 (40.42)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-39.2 to 38.3] — [estimate comment as in outcome 57, analysis 1]
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 4.7, 95% CI 2-sided [-69.4 to 78.8] — Baseline plasma HIV-1 RNA,>100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, Baseline plasma HIV-1 RNA, and treatment and Baseline plasma HIV-1 RNA interaction
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 17.4, 95% CI 2-sided [-111.1 to 145.8] — [estimate comment as in outcome 55, analysis 3]
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -1.5, 95% CI 2-sided [-37.2 to 34.1] — [estimate comment as in outcome 55, analysis 4]
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -18.0, 95% CI 2-sided [-63.2 to 27.1] — [estimate comment as in outcome 57, analysis 5]
Statistical Analysis 6: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 3.5, 95% CI 2-sided [-57.0 to 64.0] — [estimate comment as in outcome 57, analysis 6]
Statistical Analysis 7: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 95.2, 95% CI 2-sided [-14.8 to 205.2] — Age Group,>=50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 8: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 24.9, 95% CI 2-sided [-62.5 to 112.3] — [estimate comment as in outcome 55, analysis 8]
Statistical Analysis 9: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -4.2, 95% CI 2-sided [-41.5 to 33.1] — [estimate comment as in outcome 55, analysis 9]
Statistical Analysis 10: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 0.3, 95% CI 2-sided [-40.6 to 41.1] — [estimate comment as in outcome 57, analysis 10]
Statistical Analysis 11: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -51.3, 95% CI 2-sided [-163.6 to 60.9] — [estimate comment as in outcome 57, analysis 11]
Statistical Analysis 12: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Median Difference (Net) = -20.1, 95% CI 2-sided [-125.3 to 85.0] — [estimate comment as in outcome 57, analysis 12]
Statistical Analysis 13: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 66.2, 95% CI 2-sided [-43.7 to 176.2] — [estimate comment as in outcome 57, analysis 13]

59. Secondary Outcome: Change From Baseline in EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) Utility Score at Weeks 4, 24, 48
Description: EQ-5D-5L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has 1 question assessing each of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. The health state is defined by combining the levels of answers from each of the 5 questions. Each health state is referred to in terms of a 5 digit code. Health state 5 digit code is translated into utility score, which is valued up to 1 (perfect health) with lower values meaning worse state. EQ-5D-5L utility score ranges from -0.281 to 1. Higher scores indicate better health. Baseline was the latest pre-dose assessment (Day 1) and change from Baseline=post-dose value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 24, 48
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Scores on a scale
  Week 4, n=349, 348: number analyzed (Participants) | 349 | 348
  Week 4, n=349, 348 | 0.0130 (0.00362) | 0.0078 (0.00353)
  Week 24, n=352, 351: number analyzed (Participants) | 352 | 351
  Week 24, n=352, 351 | 0.0131 (0.00371) | 0.0168 (0.00333)
  Week 48, n=352, 351: number analyzed (Participants) | 352 | 351
  Week 48, n=352, 351 | 0.0134 (0.00384) | 0.0129 (0.00349)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.302, MMRM; Mean Difference (Net) = 0.0052, 95% CI 2-sided [-0.0047 to 0.0152] — Week 4. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count (factor), and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit with visit as the repeated factor
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.450, MMRM; Mean Difference (Net) = -0.0038, 95% CI 2-sided [-0.0136 to 0.0060] — Week24. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count (factor), and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit with visit as the repeated factor
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.934, MMRM; Mean Difference (Net) = 0.0004, 95% CI 2-sided [-0.0098 to 0.0106] — Week48. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count (factor), and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit with visit as the repeated factor

60. Secondary Outcome: Change From Baseline in EQ-5D-5L Utility Score at Week 96
Description: as for outcome 59
Time Frame: Baseline (Day 1) and Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 352 | 351
Scores on a scale | 0.0079 (0.00450) | 0.0091 (0.00408)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.842, MMRM; Mean Difference (Net) = -0.0012, 95% CI 2-sided [-0.0132 to 0.0107] — Week 96. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

61. Secondary Outcome: Change From Baseline in EQ-5D-5L Utility Score at Week 144
Description: as for outcome 59
Time Frame: Baseline (Day 1) and Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 352 | 351
Scores on a scale | 0.0143 (0.00388) | 0.0135 (0.00365)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.879, MMRM; Mean Difference (Net) = 0.0008, 95% CI 2-sided [-0.0097 to 0.0113] — Week 144. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

62. Secondary Outcome: Change From Baseline in EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) Thermometer Scores at Weeks 4, 24 48
Description: EQ-5D-5L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L included EQ visual Analogue scale (EQ VAS) 'Thermometer' which provided Self-rated current health status. Score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). MMRM was run on the LOCF dataset, using the observed margins (OM) option. Baseline was the latest pre-dose assessment value (Day 1) and change from Baseline=post-dose value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 24, 48
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 356 | 358
Scores on a scale
  Week 4, n=349, 348: number analyzed (Participants) | 349 | 348
  Week 4, n=349, 348 | 2.3 (0.48) | 1.2 (0.52)
  Week 24, n=352, 350: number analyzed (Participants) | 352 | 350
  Week 24, n=352, 350 | 3.7 (0.54) | 3.2 (0.51)
  Week 48, n=352, 350: number analyzed (Participants) | 352 | 350
  Week 48, n=352, 350 | 4.3 (0.49) | 2.8 (0.49)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.137, MMRM; Mean Difference (Net) = 1.1, 95% CI 2-sided [-0.3 to 2.4] — Week 4. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA (factor),Baseline CD4+ cell count (factor), Baseline EQ-5D thermometer, treatment*visit and Baseline EQ-5D thermometer*visit with visit as the repeated factor
Statistical Analysis 2: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.458, MMRM; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.9 to 2.0] — Week24. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA (factor),Baseline CD4+ cell count (factor), Baseline EQ-5D thermometer, treatment*visit and Baseline EQ-5D thermometer*visit with visit as the repeated factor
Statistical Analysis 3: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.031, MMRM; Mean Difference (Net) = 1.5, 95% CI 2-sided [0.1 to 2.8] — Week48. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA (factor),Baseline CD4+ cell count (factor), Baseline EQ-5D thermometer, treatment*visit and Baseline EQ-5D thermometer*visit with visit as the repeated factor

63. Secondary Outcome: Change From Baseline in EQ-5D-5L Thermometer Scores at Week 96
Description: EQ-5D-5L questionnaire provided a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L included EQ visual Analogue scale (EQ VAS) 'Thermometer' which provided Self-rated current health status. Score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). MMRM was run on the LOCF dataset, using the observed margins (OM) option. Baseline was the latest pre-dose assessment value (Day 1) and change from Baseline=post-dose value minus Baseline value. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC-Double Blind Phase | DTG + TDF/FTC-Double Blind Phase
Number analyzed (Participants) | 352 | 350
Scores on a scale | 4.1 (0.51) | 2.4 (0.56)
Statistical Analysis 1: Comparison: DTG + 3TC-Double Blind Phase vs DTG + TDF/FTC-Double Blind Phase; Test type: Other; p = 0.027, MMRM; Mean Difference (Net) = 1.7, 95% CI 2-sided [0.2 to 3.2] — Week 96. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

64. Secondary Outcome: Change From Baseline in EQ-5D-5L Thermometer Scores at Week 144
Description: as for outcome 63
Time Frame: Baseline (Day 1) and Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 352 | 350
Scores on a scale | 5.2 (0.48) | 3.0 (0.50)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.001, MMRM; Mean Difference (Net) = 2.3, 95% CI 2-sided [0.9 to 3.6] — Week 144. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-SAEs were collected up to Week 148 in Double-blind Phase + Open-label Phase and from Week 148 to Week 280 in Continuation Phase
Description: All-cause mortality, SAEs and non-SAEs were reported for the Safety Population for the Double-blind Phase + Open-label Phase. Safety-Continuation Population was used for the Continuation Phase which comprises all participants who received at least 1 dose of study treatment after entering the Continuation Phase
Groups:
- DTG + 3TC-Double-blind Phase + Open-label Phase: Participants received a two-drug regimen of DTG + 3TC administered orally, once daily until Week 96 in double-blind phase and participants continued to receive DTG + 3TC from Week 96 to Week 148 in the open-label phase.
- DTG + TDF/FTC-Double-blind Phase + Open-label Phase: Participants received a three-drug regimen of DTG + TDF/FTC FDC administered orally, once daily until Week 96 in double-blind phase and participants continued to receive DTG + TDF/FTC FDC from Week 96 to Week 148 in the open-label phase.
- DTG + 3TC-Continuation Phase: Participants received a DTG + 3TC administered orally, once daily from Week 148 to Week 280 in the continuation phase.
Arm/Group | DTG + 3TC-Double-blind Phase + Open-label Phase | DTG + TDF/FTC-Double-blind Phase + Open-label Phase | DTG + 3TC-Continuation Phase
All-Cause Mortality (participants affected / at risk) | 1/356 | 0/358 | 0/233
Serious Adverse Events (participants affected / at risk) | 37/356 | 38/358 | 5/233
Other Adverse Events (participants affected / at risk) | 272/356 | 268/358 | 46/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 3TC-Double-blind Phase + Open-label Phase (N=356) | DTG + TDF/FTC-Double-blind Phase + Open-label Phase (N=358) | DTG + 3TC-Continuation Phase (N=233)
Hepatitis A (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Chagoma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 3TC-Double-blind Phase + Open-label Phase (N=356) | DTG + TDF/FTC-Double-blind Phase + Open-label Phase (N=358) | DTG + 3TC-Continuation Phase (N=233)
Headache (Nervous system disorders) | 51 (80) | 47 (82) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 50 (69) | 53 (73) | 0 (0)
Nasopharyngitis (Infections and infestations) | 49 (74) | 58 (84) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 37 (50) | 33 (41) | 7 (8)
Insomnia (Psychiatric disorders) | 29 (33) | 36 (40) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (13) | 32 (37) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (31) | 25 (28) | 0 (0)
Pharyngitis (Infections and infestations) | 38 (49) | 30 (43) | 6 (8)
Syphilis (Infections and infestations) | 38 (45) | 40 (47) | 6 (6)
Bronchitis (Infections and infestations) | 30 (36) | 21 (23) | 0 (0)
Pyrexia (General disorders) | 18 (24) | 12 (13) | 0 (0)
Fatigue (General disorders) | 16 (19) | 14 (15) | 0 (0)
Influenza (Infections and infestations) | 24 (28) | 18 (20) | 0 (0)
Influenza like illness (General disorders) | 19 (20) | 16 (25) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 19 (19) | 0 (0)
Sinusitis (Infections and infestations) | 15 (17) | 15 (20) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 16 (16) | 16 (19) | 0 (0)
Gastroenteritis (Infections and infestations) | 17 (19) | 15 (15) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 17 (19) | 0 (0)
Depression (Psychiatric disorders) | 18 (20) | 17 (18) | 0 (0)
Gonorrhoea (Infections and infestations) | 16 (22) | 13 (18) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 15 (15) | 0 (0)
Tonsillitis (Infections and infestations) | 13 (15) | 12 (13) | 0 (0)
Dizziness (Nervous system disorders) | 10 (13) | 10 (10) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 22 (24) | 0 (0)
Herpes zoster (Infections and infestations) | 8 (8) | 13 (13) | 0 (0)
Hypertension (Vascular disorders) | 16 (18) | 14 (14) | 5 (9)
Dyspepsia (Gastrointestinal disorders) | 13 (20) | 12 (13) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 21 (25) | 16 (17) | 0 (0)
Anxiety (Psychiatric disorders) | 19 (24) | 15 (18) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 15 (26) | 12 (18) | 0 (0)
Respiratory tract infection (Infections and infestations) | 9 (13) | 10 (19) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 8 (10) | 9 (15) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 25 (25) | 22 (23) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6 (9) | 10 (12) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 15 (24) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (12) | 9 (10) | 0 (0)
Gastritis (Gastrointestinal disorders) | 10 (11) | 6 (6) | 0 (0)
Toothache (Gastrointestinal disorders) | 11 (15) | 9 (11) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 7 (7) | 0 (0)
Chlamydial infection (Infections and infestations) | 14 (15) | 10 (10) | 0 (0)
Urethritis (Infections and infestations) | 9 (11) | 13 (13) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (11) | 13 (13) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 8 (9) | 7 (8) | 0 (0)
Tooth infection (Infections and infestations) | 10 (10) | 7 (7) | 0 (0)
Acute sinusitis (Infections and infestations) | 4 (4) | 8 (9) | 0 (0)
Oral herpes (Infections and infestations) | 9 (11) | 8 (9) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 8 (12) | 9 (12) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 9 (16) | 5 (5) | 0 (0)
Conjunctivitis (Infections and infestations) | 8 (8) | 6 (6) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 16 (18)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (9) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (11) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 6 (6) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 5 (7) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 8 (13) | 0 (0)
Seasonal allergy (Immune system disorders) | 8 (10) | 8 (12) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (8) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 9 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT02831673/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02831673/SAP_003.pdf